Pacira Pharmaceuticals, Inc. EXPAREL

| <b>Document:</b> | Statistical Analysis Plan |
|---|---|
| Official Title: | A Phase 3, Multicenter, Randomized, Double-Blind, Parallel-Group, |
| | Placebo-Controlled Study to Assess the Efficacy and Safety of |
| | Intercostal Nerve Block with Liposome Bupivacaine in Subjects |
| | Undergoing Posterolateral Thoracotomy |
| NCT Number: | NCT01802411 |
| <b>Document Date:</b> | February 26, 2013 |



# STATISTICAL ANALYSIS PLAN

A Phase 3 Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Assess the Efficacy and Safety of Intercostal Nerve Block with Liposome Bupivacaine in Subjects Undergoing Posterolateral Thoracotomy

**Protocol No.:** 402-C-322

**IND No.:** 69,198

**Study Phase:** 3

Study Drug: Liposome Bupivacaine

Date: 26 February 2013

**Prepared by:** Janice Lookabaugh, MPH

Statistician, Consultant

**Sponsor:** Pacira Pharmaceuticals, Inc.

10450 Science Center Drive

San Diego, CA 92121

Telephone: (858) 625-2424

Fax: (858) 625-0804

### Confidentiality Statement

The information contained in this document is confidential and the property of Pacira Pharmaceuticals, Inc. It should not be reproduced, revealed, or sent to third parties other than Institutional Review Boards/Independent Ethics Committees and the Investigator's research support staff participating in the conduct of the study without the prior written authorization of Pacira Pharmaceuticals, Inc.

# SIGNATURE PAGE

| Enlower | 01 March 2013 |
|-------------------------------------------------|---------------|
| Erol Onel, MD | Date |
| Executive Medical Director | |
| $\sim M_{\odot}$ | |
| ( Jey Pater | 01 March 2013 |
| Gary Patou, MD | Date |
| Chief Medical Officer | |
| Patura mill | 01 March 2013 |
| Patricia Mills, RN | Date |
| Sr. Director, Drug Safety and Pharmacovigilance | |
| Jenice Lookaland | 01 March 2013 |
| Janice Lookabaugh, MPH | Date |
| Statistician Consultant | |

# **TABLE OF CONTENTS**

| TITLE P | AGE | 1 |
|---------|----------------------------------------------------------|----|
| SIGNAT | URE PAGE | 2 |
| TABLE ( | OF CONTENTS | 3 |
| 1. | LIST OF ABBREVIATIONS | 5 |
| 2. | INTRODUCTION | 7 |
| 3. | STUDY OBJECTIVES | 8 |
| 4. | STUDY OVERVIEW | 9 |
| 5. | DEFINITIONS | 11 |
| 6. | ANALYSIS SETS | 12 |
| 7. | STATISTICAL METHODS OF ANALYSIS | 13 |
| 7.1. | General Principles | 13 |
| 7.1.1. | Calculation of AUC of NRS | 13 |
| 7.1.2. | Imputation of NRS Pain Intensity Scores. | 14 |
| 7.1.3. | Handling Missing Values. | 15 |
| 7.1.4. | Multiplicity Adjustments | 16 |
| 7.1.5. | By-Center Analyses | 17 |
| 7.2. | Subject Disposition | 17 |
| 7.3. | Description of Demographics and Baseline Characteristics | 17 |
| 7.4. | Prior and Concomitant Medication | 17 |
| 7.5. | Measurements of Treatment Compliance | 18 |
| 7.6. | Efficacy Analysis | 18 |
| 7.6.1. | Efficacy Variables | 18 |
| 7.6.2. | Methods of Analysis | 19 |
| 7.7. | Pharmacokinetic Analyses | 23 |
| 7.7.1. | Pharmacokinetic Parameter Calculation Methods | 23 |
| 7.7.2. | Pharmacokinetic Concentrations and Variables | 24 |
| 7.8. | Safety Analyses. | 24 |
| 7.8.1. | Adverse Events | 24 |
| 7.8.2. | Laboratory Parameters | 25 |

| 7.8.3. | Vital Signs | 25 |
|--------|-----------------------------------------|----|
| 7.8.4. | Other Safety Parameters | 25 |
| 7.9. | Interim Analysis | 25 |
| 8. | SAMPLE SIZE CALCULATIONS | 26 |
| 9. | REFERENCES | 27 |
| 10. | LAYOUT OF TABLES, LISTINGS, AND FIGURES | 28 |

# 1. LIST OF ABBREVIATIONS

| AE | Adverse event |
|---|---|
| ANCOVA | Analysis of covariance |
| ASA | American Society of Anesthesiologists |
| ATC | Anatomic therapeutic chemical |
| AUC | Area under the curve |
| AUC <sub>(0-inf)</sub> | Area under the plasma concentration versus time curve from time 0 extrapolated to infinity |
| AUC <sub>(0-last)</sub> | Area under the plasma concentration versus time curve from time 0 to the last collection time after drug administration |
| BLOQ | Below the limit of quantification |
| CI | Confidence interval |
| C <sub>max</sub> | The maximum observed plasma concentration obtained directly from the experimental data without interpolation |
| %CV | Coefficient of variation |
| CRF | Case report form |
| CSR | Clinical study report |
| C <sub>(t)</sub> | Last observed quantifiable concentration |
| eCRF | Electronic case report form |
| ECG | Electrocardiogram |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| ICH | International Conference on Harmonisation |
| ICU | Intensive Care Unit |

| | T |
|---|---|
| IM | Intramuscular |
| IV | Intravenous |
| λz | Apparent terminal elimination rate constant |
| LOCF | Last observation carried forward |
| LS | Least squares |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NRS | Numeric rating scale |
| NRS-A | Numeric rating scale with activity |
| NRS-R | Numeric rating scale at rest |
| OBAS | Overall benefit of analgesia score |
| ORAE | Opioid-related adverse event |
| PCA | Patient-controlled analgesia |
| PK | Pharmacokinetic |
| РО | Oral |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SOC | System organ class |
| TEAE | Treatment-emergent adverse event |
| t <sub>last</sub> | Time to last quantifiable concentration |
| T <sub>max</sub> | Time to maximum concentration |
| t <sub>1/2</sub> | Half-life calculated from the apparent terminal elimination rate |
| WHO-DD | World Health Organization Drug Dictionary |
| wWOCF | Windowed worst observation carried forward |

### 2. INTRODUCTION

This statistical analysis plan (SAP) describes the planned statistical analysis and reporting of the clinical study 402-C-322 titled "A Phase 3, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Assess the Efficacy and Safety of Intercostal Nerve Block with Liposome Bupivacaine in Subjects Undergoing Posterolateral Thoracotomy".

The structure and content of this SAP provide sufficient detail to meet the requirements identified by the US Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonisation (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials [1]. All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association [2] and the Royal Statistical Society [3], for statistical practice.

The purposes of this SAP are to:

- Outline the types of analyses and presentations of data that will form the basis for drawing conclusions to the study objectives and hypotheses outlined in the protocol.
- Explain in detail how the data will be handled and analyzed, adhering to commonly accepted standards and practices for Good Statistical Practice.

The planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts. Also, post-hoc exploratory analyses not necessarily identified in this SAP may be performed to further examine study data. Any post-hoc, or unplanned, exploratory analyses performed will be clearly identified as such in the final CSR.

The following documents were reviewed in preparation of this SAP:

- Protocol 402-C-322 Amendment 1 issued on 23 September 2012.
- Case report forms (CRFs) for Protocol 402-C-322.
- ICH Guidance on Statistical Principles for Clinical Trials (E9).

The reader of this SAP is encouraged to also read the clinical study protocol and other identified documents for details on the planned conduct of this study. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analyses.

A separate SAP will be written for the analysis of electrocardiogram (ECG) data.

# 3. STUDY OBJECTIVES

The primary objective of this study is to evaluate the efficacy of intercostal nerve block using liposome bupivacaine compared with placebo in subjects undergoing posterolateral thoracotomy.

The secondary objectives are to evaluate additional efficacy parameters, assess the pharmacokinetic (PK) profile of liposome bupivacaine when administered as an intercostal nerve block, and further characterize the safety profile of liposome bupivacaine.

### 4. STUDY OVERVIEW

This is a Phase 3, multicenter, randomized, double-blind, parallel-group, placebo-controlled study in subjects undergoing posterolateral thoracotomy.

After completing screening procedures, eligible subjects will be randomized 1:1 to receive either liposome bupivacaine or placebo. Study drug will be administered after the posterolateral thoracotomy is completed (i.e., just prior to the surgical site closure).

All subjects will be required to remain in the study site for a minimum of 72 hours after the end of surgery for postsurgical assessments.

# **Postsurgical Rescue Medication**

Rescue medication should only be provided upon subject request, as needed.

#### First Rescue Medication

The first rescue medication will be intravenous (IV) fentanyl 100 mcg, which will be administered once via bolus only.

# Second Rescue Medication

For the US sites only, the second rescue medication will be a patient-controlled analgesia (PCA) pump administered opioid (morphine or hydromorphone). The PCA pump will be programmed to deliver either of the following recommended doses: (1) on-demand morphine boluses of 1.5 mg with a lockout interval of 6 minutes and an initial maximum hourly dose of 15 mg or (2) on-demand hydromorphone boluses of 0.2 mg with a lockout interval of 10 minutes and an initial maximum hourly dose of 1.2 mg. The recommended bolus doses may be adjusted according to local hospital practice; however, adding a basal rate is prohibited.

<u>For the European sites only,</u> the second rescue medication will be intramuscular (IM) administered opioid (morphine) up to 10 mg every 4 hours.

At all sites, once a subject is tolerating oral (PO) medication, PO immediate-release oxycodone may be administered, as needed (but not more than 10 mg every 4 hours).

Subjects who do not achieve adequate pain relief with this regimen will be withdrawn from the study and followed for safety only.

## **Postsurgical Assessments**

Subjects will be evaluated for pain using the numeric rating scale (NRS) at rest (NRS-R) at baseline and 1, 2, 4, 8, 12, 24, 36, 48, 60, and 72 hours following surgery, at first request for rescue pain medication, and on Day 12. Subjects will also be evaluated for pain with activity using the NRS with activity (NRS-A) at baseline, and 24, 48, and 72 hours following surgery and on Day 12.

Neurological assessments will be conducted at baseline, 15 minutes, 30 minutes, and 1, 2, 4, 8, 12, 18, 24, 30, 36, 42, 48, 60, and 72 hours after surgery. The cardiac assessment (i.e., ECG

recordings) will be started at baseline (approximately 1 hour prior to surgery) and continue for a total of 72 hours. The sensory function assessment (i.e., cold test) will be conducted at baseline, when the subject wakes up after surgery, and at 2, 4, 12, 24, 36, 48, 60, and 72 hours after surgery, or until the subject's sensitivity to cold has returned in two consecutive evaluations.

The overall benefit of analgesia score (OBAS) questionnaire will be completed at 24, 48, and 72 hours following surgery. The subject's overall satisfaction with postsurgical pain control will be assessed 72 hours following surgery, on Day 12, and on Day 30 using a 5-point Likert scale. A wound healing assessment will be performed by the physician on Day 12. Predefined, treatment-emergent opioid-related adverse events (AEs) will be assessed at 72 hours following surgery. Adverse events will be recorded through the Day 30 follow-up contact.

### **Pharmacokinetic Assessments**

Blood samples for PK analysis will be obtained from subjects at specific sites at baseline, 15 minutes, 30 minutes, and 1, 2, 4, 8, 12, 24, 36, 48, 60, and 72 hours after the end surgery.

Unscheduled blood samples also may be collected if a cardiac or neurological event occurs that the Investigator believes may be associated with high levels of systemic bupivacaine.

# 5. **DEFINITIONS**

The terms "study site" and "center" are used interchangeably.

Time 0 is defined as the start time of study drug administration for the PK analyses, and as the end time of surgery for the efficacy analyses.

Study day: Day 1 is defined as the day study drug is administered. Positive study days will be measured forward in time from Day 1, with Day 2 being the calendar day immediately following the day study drug is administered. Day -1 is the calendar day immediately preceding the day study drug is administered and negative study days will be measured backward from Day -1.

Study visits and time points will be determined from the scheduled times as reported on the electronic CRFs (eCRFs) for the summarization and analysis of data that are shown by time point, unless otherwise specified.

# 6. ANALYSIS SETS

The safety analysis set will include all subjects who receive study drug and will be based on actual treatment received.

The efficacy analysis set will include all subjects in the safety analysis set and will be based on randomized treatment, regardless of actual treatment received.

The PK analysis set will include all subjects in the safety analysis set who receive liposome bupivacaine and who provide sufficient samples to allow for calculation of the PK parameters required for analysis.

### 7. STATISTICAL METHODS OF ANALYSIS

# 7.1. General Principles

Descriptive statistics (the number of subjects [n], mean, standard deviation [SD], median, minimum, and maximum) will be used to summarize continuous variables. Means and medians will be presented to one more decimal place than the recorded data. Standard deviations will be presented to two more decimal places than the recorded data. Minimum and maximum values will be presented using the same number of decimal places as the recorded data. Percentages will be presented to one decimal place.

In addition, for PK parameters, geometric means and between-subject coefficient of variations (%CV) will be presented.

Frequency distributions (number [n] and percentage of subjects [%]) will be used to summarize categorical or qualitative variables. In general, the denominator for the percentage calculation will be based upon the total number of subjects in the study population for the treatment groups, unless otherwise specified.

All statistical tests will be performed against a two-sided alternative hypothesis with a significance level of 5% ( $\alpha$  = 0.05), and all confidence intervals (CIs) calculated will be two-sided 95% CIs. All tests will be declared to be statistically significant if the calculated p-value is  $\leq$  0.05 unless specified otherwise. Tests for binomial proportions will be conducted (1) using a normal approximation whenever each classification cell for each group to be compared contains expected cell counts of 5 or more subjects, or (2) using an exact method whenever any one classification cell for any one group to be compared contains expected cell counts of fewer than 5 subjects.

All analyses will be performed using SAS® software Version 9.2 or later.

Pharmacokinetic parameters will be derived using noncompartmental methods with WinNonlin® Professional Version 5.2 or later.

For the listings subjects will be listed under their randomized treatment, regardless of actual treatment received. Subjects who are randomized but do not receive study drug will be included in the listings with the treatment group identified as "Liposome bupivacaine 266 mg, Not Treated" or "Placebo, Not Treated", depending on their randomized treatment.

### 7.1.1. Calculation of AUC of NRS

Area under the curve (AUC) will be calculated using the trapezoidal method with the actual NRS pain intensity scores reported by the subject. Missing values will be imputed as described in Section 7.1.2. The time points "Baseline" and "First Rescue" will not be included in the calculation of AUC. However, "First Rescue" might be used for imputation purposes as

described in Section 7.1.2. Time 0 NRS score will be set to a score of 0. Actual times, not scheduled times, when available will be used in the calculations. Linear interpolation will be used to calculate the pain intensity score at the end of an interval. For 72 hours, as an example, if the actual time is prior to 72 hours post-dose then the actual time and the reported score will be used. In addition, the reported score will be carried forward to 72 hours. If the actual time is after 72 hours then linear interpolation between the 60-hour and 72-hour scores will be used to calculate the score at 72 hours and the time will be set to 72.

## 7.1.2. Imputation of NRS Pain Intensity Scores

For calculation of AUC of NRS pain intensity scores, the windowed worst observation carried forward (wWOCF) and last observation carried forward (LOCF) imputation procedure will be used as follows:

a) Windowed worst observation carried forward for rescue medications

For subjects who take a rescue medication, (either a per-protocol opioid or a non-per protocol opioid) or a non-opioid analgesic postsurgically, their NRS scores recorded within the window of controlled type of rescue medication (see the table below for the windows for the per-protocol rescue medications) will be replaced by the 'worst' observation. The worst observation will be the highest score in the time interval from Time 0 to up to the time prior to taking the first rescue medication. The NRS score at the first rescue will be included in this calculation. Note that NRS scores in the window that are higher than the worst value prior to rescue medication will not be overwritten. If no NRS score is available prior to the first rescue the worst observation from all available NRS scores from the subject will be used instead.

| Medication | Route | Window Used to Impute NRS |
|---------------|-------|---------------------------|
| Fentanyl | IV | 6 hours |
| Oxycodone | PO | 6 hours |
| Morphine | IV | 4 hours |
| Hydromorphone | IV | 2 hours |

IV = intravenous; NRS = numeric rating scale; PO = oral.

If non-per protocol rescue medications are given then the window will be determined post-hoc prior to breaking the blind. For non-opioid analgesics the half-life of the analgesic, if known, will be used for the window.

- b) Missing scores before the first non-missing score will be replaced by the median score at the missing time point from the other subjects in the same treatment group.
- c) Missing scores after the last non-missing score will be replaced by the LOCF.
- d) Missing scores between two non-missing scores will not be replaced (i.e., linear interpolation will be used).

e) Subjects who have no pain intensity scores recorded after surgery will have the missing scores replaced by the median score at each time point from all subjects in the same treatment group.

# 7.1.3. Handling Missing Values

### Surgery Date or Time

It is expected that all necessary information on surgery (start and stop date and time) and postsurgical rescue medication (start dates and times, doses, frequency) will be complete. Any such information that is missing and cannot be obtained through query resolution may be imputed, on a case-by-case basis, in a conservative manner that minimizes bias. For example, if pain medication taken on Day 1 has no time of administration recorded, the imputed time will be the end of surgery.

#### Rescue Pain Medication

For calculation of the total rescue pain medication usage (morphine equivalent) through a time point, if a subject is discontinued early (e.g., dies, withdraws consent, is withdrawn from the study, or is lost to follow-up) before the end of the time interval (e.g., 24 hours after study drug administration), his or her total rescue pain medication usage through the time interval will be a projected amount. For example, if a subject discontinues early at 6 hours after surgery, the projected amounts through 24 hours will be actual amount + average amount (actual amount/6 hours) multiplied by the number of hours remaining in the time interval (24-6).

#### Adverse Event or Concomitant Medications Dates or Times

For AEs or concomitant medications with missing or partially missing start/stop date/time, the following imputation rules will be applied:

### For partial start date/time:

- If the year is unknown, then the date will not be imputed and will be assigned a missing value.
- If the month is unknown, then:
  - i) If the year matches the year of the dose of study drug date, then the month and day of the dose of study drug date will be imputed.
  - ii) Otherwise, 'January' will be assigned.
- If the day is unknown, then:
  - i) If the month and year match the month and year of the dose of study drug date, then the day of the dose of study drug date will be imputed.
  - ii) Otherwise, '01' will be assigned.
- If the time is unknown, then:

- i) If the date (day, month, and year) matches the date of the administration of study drug, then the time of the dose of study drug time will be imputed.
- ii) Otherwise, "00' will be assigned.

### For partial stop date/time:

- If the year is unknown, then the date will not be imputed and will be assigned a missing value.
- If the month is unknown, then 'December' will be assigned.
- If the day is unknown, then the last day of the month will be assigned.
- If the time is unknown, then the last time of the day will be assigned (23:59).

If the above rules for stop dates result in an illogical date with regards to the dates the subject is in the study, then the stop date will be replaced with the subject's date of completion/withdrawal. Further, should the above rules not result in the most conservative date, then the imputed value may be replaced by a date that will lead to a more conservative analysis. Should this situation arise, specific details will be provided in the derived dataset specification documentation or documented in the derived analysis data set program using comments.

## Adverse Event Severity or Relationship to Study Drug

If severity of an AE is not reported, then for tables of AEs by severity, the event will be classified as 'Severe'. If relationship to study drug is not reported for an AE, then for tables of study-drug related AEs, the event will be classified as related.

### Time to Event

For calculating time to an event when only the hour, and not the minutes, is reported for the time of the event, then the minutes will be set to zero.

### 7.1.4. Multiplicity Adjustments

Since no multiple comparisons of the primary efficacy variable will be made, no alphaadjustments will be made.

Also, since there is only one primary efficacy variable and all other efficacy variables are considered secondary, no alpha-adjustments for the primary response variable will be made.

There are two secondary efficacy variables that will be analyzed using a hierarchical fixed-sequence stepwise testing procedure (see Section 7.6.1). To protect the Type 1 error rate, the testing will be performed in a sequentially rejective fashion. First, the total postsurgical opioid consumption through 72 hours will be tested. If the test of opioid consumption is significant at the two-sided 0.05 level then, and only then, the time to first opioid rescue will be tested. Each test will be declared positive at the two-sided 0.05 significance level.

# 7.1.5. By-Center Analyses

Up to 30 sites/centers in the US and Europe will enroll subjects in this study. The primary efficacy results will be summarized by site and region (US and Europe) but site will not be included in any models. Region will be included in the models.

# 7.2. Subject Disposition

The number and percentage of subjects who are in each analysis set, who completed the study, and who discontinued early from the study, along with reasons for early withdrawal, will be summarized by treatment group and for all subjects. In addition, the same summary will be produced by site and region.

# 7.3. Description of Demographics and Baseline Characteristics

Demographics and baseline characteristics will be summarized by treatment group and for all subjects for the safety analysis set. The variables to be included in the summary are age, gender, ethnicity, race, American Society of Anesthesiologists (ASA) physical status class, height (cm), and weight (kg).

Conversions between units for height and weight will use the following formulas:

Weight (kg) = weight (lb) / 2.2046226

Height (cm) = height (in) / 2.54.

If any subjects are randomized to the liposome bupivacaine group and receive placebo or any subjects are randomized to the placebo group and receive liposome bupivacaine then a similar table will be created using the efficacy analysis set.

#### 7.4. Prior and Concomitant Medications

Prior and concomitant medications will be coded using the World Health Organization Drug Dictionary (WHO-DD) and will be classified according to the default anatomical therapeutic chemical (ATC) classification system code and preferred term.

Prior medications are defined as medications with a stop date/time prior to study drug administration. Concomitant medications are defined as medications taken after the start of study drug administration (i.e., started prior to the start of study drug administration and continued after or started after the start of study drug administration).

Prior and concomitant medications will be summarized using n (%) of subjects by treatment group and for all subjects and by ATC class and preferred term for the safety analysis set. Subjects may have more than one medication per ATC category and preferred term. At each level of subject summarization, a subject will be counted once if he/she reports one or more medications at that level.

The tables of concomitant medications will not include protocol-specified rescue pain medications.

# 7.5. Measurements of Treatment Compliance

Study drug administration will be summarized by treatment group for the safety analysis set. The variables to be included are duration of injection and volume of study drug administered. Surgery will be summarized by treatment group for the efficacy analysis set. The variables to be included in the summary are length of surgery (end time minus start time, in minutes), level of index nerve injected, length of time in the Intensive Care Unit (ICU) (hours), and number and percentage of subjects with at least one chest tube and length of time from end of surgery to removal of last chest tube, for subjects who have a chest tube inserted.

# 7.6. Efficacy Analysis

All summaries of the efficacy variables will use the efficacy analysis set, which will be based on randomized treatment.

# 7.6.1. Efficacy Variables

The primary efficacy variable is the AUC of the NRS-R pain intensity scores through 72 hours.

The secondary efficacy variables are:

- Total postsurgical opioid consumption (in mg) through 72 hours.
- Time to first opioid rescue.

The tertiary efficacy variables are (the order of these variables has been changed from the order in the protocol to reflect how they will be discussed in the CSR):

- The NRS-R and NRS-A pain intensity scores at each assessed time point.
- The AUC of the NRS-R pain intensity scores through 24, 36, 48, and 60 hours.
- The AUC of the NRS-R pain intensity scores from 24-48 and 48-72 hours.
- Proportion of subjects who are pain free (defined as an NRS pain intensity score of 0 or 1) at each assessed time point.
- Total postsurgical opioid consumption (in mg) through 24, 36, 48, and 60 hours.
- Proportion of subjects who receive the following rescue medication(s):
  - o Subjects who receive no rescue medication.
  - o Subjects who only receive IV fentanyl as a rescue medication.
  - o Subjects who receive IV fentanyl and a second opioid medication.
- Overall benefit of analgesia score questionnaire at 24, 48, and 72 hours.

- Subject satisfaction with postsurgical pain control at 72 hours, Day 12, and Day 30.
- Time to sensitivity to cold (listed in the protocol as "Proportion of subjects at each time point with sensitivity to cold anywhere within the dermatomes supplied by any of the nerves to which study drug was administered").
- Incidence of predefined treatment-emergent opioid-related AEs (ORAEs) (diffuse pruritus, overt respiratory depression, urinary retention as measured by need for postsurgical bladder catheterization, constipation, sedation, confusion, delirium, vomiting, or need for antiemetic medication) at 72 hours.

# 7.6.2. Methods of Analysis

### 7.6.2.1 Primary Efficacy Variable

The primary efficacy variable is the AUC of the NRS-R pain intensity scores through 72 hours calculated using the wWOCF + LOCF imputation method described in Section 7.1.2.

Liposome bupivacaine will be compared to placebo using analysis of covariance (ANCOVA) with treatment and region (US and Europe) as main effects and the baseline NRS-R pain intensity score as a covariate. Based on the model, the least squares (LS) means, LS mean difference between the two treatment groups, 95% CI for the LS mean difference(s) between liposome bupivacaine and placebo, and p-value will be reported.

Descriptive statistics of the primary efficacy variable will also be shown by region and site.

# 7.6.2.2 Secondary Efficacy Variables

The secondary efficacy variables for this study are:

- Total postsurgical opioid consumption through 72 hours.
- Time to first opioid rescue.

For total postsurgical opioid consumption, opioid medications will be converted to a morphine equivalent amount (see the table below). The converted amounts will be totaled for each subject and used in the analysis. Projected amounts, for subjects who discontinue early, will be calculated as described in Section 7.1.3.

| Medication | Unit | Route | Conversion (Multiplication)<br>Factor |
|---------------|------|----------|---------------------------------------|
| Fentanyl | mcg | IV | 0.1 |
| Oxycodone | mg | РО | 0.5 |
| Morphine | mg | IV or IM | 1 |
| Hydromorphone | mg | IV | 6.7 |

IV = intravenous; PO = oral.

If any other opioids are administered, then the conversion factor will be determined post-hoc prior to breaking the blind.

Prior to analysis, the natural logarithm transformation will be applied to the total amount. When total amount of opioids used is 0, the result will be changed to the lesser of 1 or 0.5 of the smallest total amount observed in the study prior to being transformed with the natural logarithm. To test for significant differences between liposome bupivacaine and placebo, an analysis of variance (ANOVA) with treatment and region (US and Europe) as main effects will be used. Based on the model, the geometric LS means, geometric LS mean ratio of liposome bupivacaine to placebo, 95% CI for the geometric LS mean ratio of liposome bupivacaine to placebo, and p-value will be reported.

For the analysis of time to first opioid rescue, time to first opioid rescue will be computed in hours as the date/time of the first opioid rescue minus the date/time of the end of surgery. If a subject is not administered an opioid, the time to first administration will be censored at 72 hours after surgery or at the time of last follow-up, whichever is earliest. Time of last follow-up will be defined as the later of (1) the last pain assessment, (2) the start time of the last rescue or concomitant medication, or (3) the start time of the last AE.

Time to first opioid rescue will be analyzed by the Kaplan-Meier method. The n (%) of subjects administered an opioid as well as the n (%) of censored observations will be presented for each treatment group. In addition, Kaplan-Meier estimates in terms of the median and its 95% CI, and the 25<sup>th</sup> and 75<sup>th</sup> percentiles will be presented for each treatment. A Log-rank test with region (US and Europe) as a stratifying variable will be used to compare liposome bupivacaine to placebo.

The secondary efficacy measures will be analyzed using a hierarchical fixed-sequence stepwise testing procedure. To protect the Type 1 error rate, the testing will be performed in a sequentially rejective fashion. First, the total postsurgical opioid consumption through 72 hours will be tested. If the test of opioid consumption is significant at the two-sided 0.05 level then, and only then, the time to first opioid rescue will be tested. Each test will be declared positive at the two-sided 0.05 significance level.

# 7.6.2.3 Tertiary Efficacy Variables

The following describes the statistical analyses to be performed.

# NRS-R, NRS-A, and AUC of the NRS-R Pain Intensity Scores

For the tertiary efficacy variables NRS-R, NRS-A, and the AUC of the NRS-R pain intensity scores, the same analyses as those for the primary efficacy variable will be performed, except that the baseline NRS-A score will be used as the covariate for all variables using the NRS-A.

# Proportion of Subjects Who are Pain Free

'Pain free' is defined as an NRS-R pain intensity score of 0 or 1. The number and percentage of subjects who are pain free will be summarized by treatment group for each time point. A chi-square test will be used to compare liposome bupivacaine to placebo.

# Total Postsurgical Opioid Consumption Through 24, 36, 48, and 60 Hours

For the tertiary efficacy variable of total opioid consumption through each of the time periods, the same analysis as that for the secondary efficacy variable of total opioid consumption through 72 hours will be performed.

# Subjects Who Receive Rescue Medication

The category of 'Subjects who received no rescue medication' is defined as subjects who did not receive any medication reported on the three Rescue Medication eCRFs.

The category of 'Subjects who only received IV fentanyl as a rescue medication' is defined as subjects who received IV fentanyl based on the First Rescue Medication eCRF and did not receive any medication based on all of the Second Rescue Medication eCRFs.

The category of 'Subjects who received IV fentanyl and a second opioid medication' is defined as subjects who received IV fentanyl based on the First Rescue Medication eCRF and who either received a medication based on any of the Second Rescue Medication eCRFs or reported an opioid on the Concomitant Medications eCRF (with a start date within 72 hours of the end of surgery).

The number and percentage of subjects who are in each of the above categories will be summarized by treatment group. A chi-square test will be used to compare liposome bupivacaine to placebo for each of the categories.

#### Overall Benefit of Analgesia Score Questionnaire

The OBAS is calculated as follows:

- 1. Add all of the scores of questions one to six.
- 2. To this number, add four.
- 3. Subtract the score of question seven from this number.

Summary statistics will be provided by treatment group at each time point. A Wilcoxon Rank Sum test will be used to compare liposome bupivacaine to placebo.

### Subject Satisfaction with Postsurgical Pain Control

Subjects will rate their satisfaction with postsurgical pain control as 'Extremely dissatisfied', 'Dissatisfied', 'Neither satisfied nor dissatisfied', 'Satisfied', or 'Extremely satisfied' at 72 hours and on Day 30. The categories will be summarized by treatment group at each time point. A Wilcoxon Rank Sum test will be used to compare liposome bupivacaine to placebo.

### Time to Sensitivity to Cold

Once a subject reports sensitivity to cold on two consecutive evaluations the subject will no longer be tested. The time to sensitivity to cold will be defined as the time of the first of two consecutive evaluations when the subject reports sensitivity to cold. Time to sensitivity to cold will be calculated from the end of surgery. If a subject never reports sensitivity to cold or never reports sensitivity to cold on two consecutive evaluations then the time will be censored at 72 hours after the end of surgery or at the time of the last follow-up, whichever is earliest. Time of last follow-up will be defined as the later of (1) the last pain assessment, (2) the start time of the last rescue or concomitant medication, or (3) the start time of the last AE.

Time to sensitivity to cold will be analyzed by the Kaplan-Meier method. The n (%) of subjects with sensitivity to cold as well as the n (%) of censored observations will be presented for each treatment group. In addition, Kaplan-Meier estimates in terms of the median and its 95% CI, and the 25<sup>th</sup> and 75<sup>th</sup> percentiles will be presented for each treatment group. A log-rank test will be used to compare liposome bupivacaine to placebo.

# <u>Incidence of Predefined Treatment-Emergent Opioid-Related Adverse Events</u>

The determination of whether a subject had a treatment-emergent ORAE will be based solely on responses on the Predefined Treatment-Emergent ORAEs eCRF. The number and percentage of subjects who have at least one ORAE will be summarized by treatment group. A chi-square test will be used to compare liposome bupivacaine to placebo.

The number and percentage of subjects who have each of the individual ORAEs will also be summarized by treatment group, although no statistical tests will be performed.

# 7.7. Pharmacokinetic Analyses

#### 7.7.1. Pharmacokinetic Parameter Calculation Methods

Pharmacokinetic parameters will be calculated by noncompartmental analysis method from concentration-time data using WinNonlin Professional following these guidelines:

- Actual sampling times relative to study drug administration will be used for all calculations of the PK parameters. If there is any doubt as to the actual time a sample was taken, then the scheduled time will be used. Descriptive statistics will be used to summarize the PK parameters.
- There will be no imputation of missing data.

For the calculation of AUCs from PK concentrations, concentration below the limit of quantification (BLOQ) will be handled as follows:

- Pre-dose values will be set to zero.
- All remaining BLOQ values will be set to missing.

Pharmacokinetic parameters will be estimated according to the following guidelines:

- The maximum observed plasma concentration (C<sub>max</sub>) will be obtained directly from the concentration-time data.
- Time to maximum concentration  $(T_{max})$  is the time at which  $C_{max}$  is observed.
- The apparent terminal elimination rate constant ( $\lambda_Z$ ) will be estimated at terminal phase by linear regression after log-transformation of the concentrations:
  - Only those data points that are judged to describe the terminal log-linear decline will be used in the regression.
  - A minimum number of three data points in the terminal phase will be used in calculating  $\lambda_z$  with the line of regression starting at any post- $C_{max}$  data point ( $C_{max}$  should not be part of the regression slope) and including the last observed quantifiable concentration ( $C_{(t)}$ ) and the time to last quantifiable concentration ( $t_{last}$ ).
  - The adjusted correlation coefficient (R<sup>2</sup> adjusted) in general should be greater than 0.90. Any value less than 0.90 may be used at the pharmacokineticist's best knowledge and judgment.
  - An appropriate number of decimal places should be used for  $\lambda_z$  to enable the reported value of half-life ( $t_{1/2}$ ) to be calculated.
- Half-life  $(t_{1/2})$  will be calculated as  $\ln 2/\lambda_z$ .

- The AUC will be calculated as follows:
  - The linear trapezoidal method will be employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method will be used for those arising from decreasing concentrations.
  - AUC<sub>(0-t)</sub> =  $\int_0^t \mathbf{C}(\mathbf{t}) d\mathbf{t}$ .
  - $AUC_{(0-inf)} = \int_0^t \mathbf{C}(\mathbf{t}) d\mathbf{t} + \int_{\mathbf{t}}^{\infty} \mathbf{C}(\mathbf{t}) d\mathbf{t} = AUC_{(0-t)} + C_t/\lambda_{z}$
  - C<sub>(t)</sub> is last observed quantifiable concentration.

#### 7.7.2. Pharmacokinetic Concentrations and Variables

The analysis of the PK data will be based on the PK analysis set. Only data from the subjects in the liposome bupivacaine treatment group will be presented in the summary tables and listings.

Bupivacaine plasma concentrations will be listed by subject, nominal time, and actual time. Concentrations that are BLOQ will be indicated by BLOQ in this listing.

Plasma concentrations will be summarized at each time point. The following descriptive statistics will be presented for plasma concentrations obtained at each nominal time point: n, geometric mean, arithmetic mean, SD, %CV, minimum, median, and maximum.

Pharmacokinetic parameters will be summarized. Descriptive statistics for calculated PK parameters will include: n, arithmetic mean, SD, %CV, geometric mean, median, minimum and maximum values. Geometric mean will not be presented for  $T_{max}$ . Values of %AUC extrapolated > 20% will be flagged in the listings.

Individual plasma concentration versus actual times will be plotted in linear and semi-logarithmic scale.

# 7.8. Safety Analyses.

All summaries of the safety data will use the safety analysis set.

#### 7.8.1. Adverse Events

All AEs will be coded and summarized by system organ class (SOC) and preferred term based on the Medical Dictionary for Regulatory Activities (MedDRA) coding dictionary.

An AE will be considered treatment-emergent if the onset is any time on or after study drug administration through Day 30.

Only treatment-emergent AEs (TEAEs) that were not solicited from the Neurological Assessment or from the Opioid-Related Adverse Event Questionnaire will be summarized in the tables. All other AEs, those that occur after randomization but prior to study drug

administration, AEs that occur after Day 30, or AEs that were solicited from the Neurological Assessment or from the Opioid-Related Adverse Event Questionnaire will appear in listings only.

Treatment-emergent AEs will be summarized [n (%)] and grouped by SOC and preferred term for each treatment group and for all subjects. If a subject experiences more than one episode of a particular TEAE, the subject will be counted only once for that event at each level of summarization (overall, by SOC, and by preferred term).

Similarly, TEAEs will be summarized in terms of maximum severity ('Mild', 'Moderate', and 'Severe'), study drug-related TEAEs, and serious AEs.

## 7.8.2. Laboratory Parameters

Not applicable.

# 7.8.3. Vital Signs

Descriptive summaries of actual value and changes from Baseline will be calculated for systolic blood pressure, diastolic blood pressure, and heart rate.

### 7.8.4. Other Safety Parameters

## Neurological Assessments

The proportion of subjects who are oriented will be summarized by treatment group at each time point. Subjects who were 'not assessable' will not be included in the calculation of the proportion. The proportion of subjects who have at least one of the neurological events and the proportion of subjects who have each of the neurologic events will be summarized by treatment group.

### Physician's Satisfaction with Wound Healing

The physician's satisfaction with wound healing will be assessed as 'Extremely dissatisfied', 'Dissatisfied', 'Neither satisfied nor dissatisfied', 'Satisfied', or 'Extremely satisfied' on Day 30. The categories will be summarized by treatment group at each time point. A Wilcoxon Rank Sum test will be used to compare liposome bupivacaine to placebo.

# 7.9. Interim Analysis

No interim analyses are planned.

# 8. SAMPLE SIZE CALCULATIONS

A study population of approximately 180 subjects is planned with approximately 90 subjects in each treatment group (liposome bupivacaine and placebo). The sample size was estimated based on the results of a Phase 3 wound infiltration hemorrhoidectomy study of liposome bupivacaine versus placebo where the mean (SD) AUC of the NRS-R pain intensity scores through 72 hours was 141 (101) and 202 (104) for the liposome bupivacaine and placebo groups, respectively. A two-group t-test with 0.05 two-sided significance level will have > 97% power to detect a difference in means of 61, assuming that the common SD is 104, when the sample size in each group is 90.

# 9. **REFERENCES**

- 1. US Federal Register. International Conference on Harmonisation; Guidance on Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration [Docket No. 97D-0174]. Federal Register Volume 63, Number 179, pages 49583-49598. 16 September 1998.
- 2. American Statistical Association. Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, 07 August 1999. <a href="http://www.amstat.org/profession/ethicalstatistics.html">http://www.amstat.org/profession/ethicalstatistics.html</a>
- 3. Royal Statistical Society. The Royal Statistical Society: Code of Conduct, August 1993. <a href="http://www.rss.org.uk/about/conduct.html">http://www.rss.org.uk/about/conduct.html</a>.

# 10. LAYOUT OF TABLES, LISTINGS, AND FIGURES

The following are planned summary tables for Protocol 402-C-322. Tables will be numbered according to the nomenclature used to support the CSR. The final table numbering may be different from the SAP. No amendment will be made for changes in table numbering. All headers, titles, footnotes, and footers specified in the table templates will be displayed in the produced output unless otherwise specified. Notes to programmers will not be included in the tables. There will be a footnote in all tables that includes the program name, SAS version number, and the date that the output was produced.

#### **Planned Tables**

| Table | |
|---|---|
| Number | Table Title |
| | Subject Disposition |
| 14.1.1.1 | (All Subjects) |
| | Subject Disposition by Region and Site |
| 14.1.1.2 | (All Subjects) |
| | Demographic and Baseline Characteristics |
| 14.1.2 | (Safety Analysis Set) |
| | Prior Medications |
| 14.1.3.1 | (Safety Analysis Set) |
| | Concomitant Medications |
| 14.1.3.2 | (Safety Analysis Set) |
| | Study Drug Administration |
| 14.2.1.1 | (SafetyAnalysis Set) |
| | Surgery |
| 14.2.1.2 | (Efficacy Analysis Set) |
| | AUC of NRS-R Pain Intensity Scores Through 72 Hours |
| | wWOCF + LOCF Imputation for the Pain Scores |
| 14.2.2.1.1 | (Efficacy Analysis Set) |
| | AUC of NRS-R Pain Intensity Scores Through 72 Hours by Region and |
| | Site |
| | wWOCF + LOCF Imputation for the Pain Scores |
| 14.2.2.1.2 | (Efficacy Analysis Set) |
| | Total Postoperative Consumption (mg) of Opioid Rescue Pain Medication |
| | Through 72 Hours |
| 14.2.2.2 | (Efficacy Analysis Set) |

# **Planned Tables Continued**

| Table | |
|---|---|
| Number | Table Title |
| Titalinger | Time to First Opioid Rescue |
| 14.2.2.3.2 | (Efficacy Analysis Set) |
| | NRS-R Pain Intensity Scores |
| 14.2.2.4 | (Efficacy Analysis Set) |
| | NRS-A Pain Intensity Scores |
| 14.2.2.5 | (Efficacy Analysis Set) |
| | AUC of NRS-R Pain Intensity Scores Through 24, 36, 48, and 60 Hours |
| | wWOCF + LOCF Imputation for the Pain Scores |
| 14.2.2.6 | (Efficacy Analysis Set) |
| | AUC of NRS-R Pain Intensity Scores 24-48 and 48-72 Hours |
| | wWOCF + LOCF Imputation for the Pain Scores |
| 14.2.2.7 | (Efficacy Analysis Set) |
| | Percentage of Subjects who are Pain Free at Each Time Point |
| 14.2.2.8 | (Efficacy Analysis Set) |
| | Total Postoperative Consumption (mg) of Opioid Rescue Pain Medication |
| | Through 24, 36, 48, and 60 Hours |
| 14.2.2.9 | (Efficacy Analysis Set) |
| | Subjects who Received Rescue Medication Through 72 Hours |
| 14.2.2.10 | (Efficacy Analysis Set) |
| | Overall Benefit of Analgesia Score Questionnaire (Total Scores) |
| 14.2.2.11 | (Efficacy Analysis Set) |
| | Subject Satisfaction with Postsurgical Pain Control |
| 14.2.2.12 | (Efficacy Analysis Set) |
| | Time to Sensitivity to Cold |
| 14.2.2.13 | (Efficacy Analysis Set) |
| | Incidence of Predefined Treatment-Emergent Opioid-Related Adverse |
| | Events |
| 14.2.2.14 | (Efficacy Analysis Set) |
| | Bupivacaine Plasma Concentrations (ng/mL) |
| | Study Part 1 |
| 14.2.3.1 | (PK Analysis Set) |
| | Bupivacaine Plasma Pharmacokinetic Parameters |
| 14.2.3.2 | Study Part 1 (PK Analysis Set) |
| 14.2.3.2 | Overview of Treatment-Emergent Adverse Events |
| 14.3.1.1 | (Safety Analysis Set) |
| 14.5.1.1 | Incidence of Treatment-Emergent Adverse Events |
| 14.3.1.2 | (Safety Analysis Set) |
| 17.3.1.4 | Incidence of Study Drug Related Treatment-Emergent Adverse Events |
| 14.3.1.3 | (Safety Analysis Set) |
| 17.3.1.3 | (Sairty Allalysis Sti) |

# **Planned Tables Continued**

| Table | |
|----------|------------------------------------------------------------|
| Number | Table Title |
| | Incidence of Treatment-Emergent Adverse Events by Severity |
| 14.3.1.4 | (Safety Analysis Set) |
| | Incidence of Serious Treatment-Emergent Adverse Events |
| 14.3.1.5 | (Safety Analysis Set) |
| | Vital Signs |
| 14.3.2.1 | (Safety Analysis Set) |
| | Vital Signs Change from Baseline |
| 14.3.2.2 | (Safety Analysis Set) |
| | Neurological Assessment |
| 14.3.3 | (Safety Analysis Set) |
| | Physician Satisfaction with Wound Healing |
| 14.3.4 | (Safety Analysis Set) |

# **Planned Listings**

| Listing | |
|---|---|
| Number | Listing Title |
| 16.1.1 | Eligibility |
| 16.1.2 | Unblinding |
| 16.1.3 | Subject Populations and Discontinuations |
| 16.1.4 | Hospital Discharge |
| 16.2 | Demographics and Baseline Characteristics |
| 16.3.1 | Medical History |
| 16.3.2 | Physical Examination |
| 16.3.3 | Electrocardiogram Recording (Holter Monitoring) |
| | Prior and Concomitant Medications (Except for Protocol-Defined Rescue |
| 16.3.4 | Pain Medications) |
| 16.4.1 | Study Drug Exposure |
| 16.4.2 | Surgery |
| 16.4.3 | Intensive Care Unit and Chest Tube Removal |
| 16.5.1.1 | Pain Intensity Scores at Rest and with Activity |
| | AUC of NRS-R Pain Intensity Scores |
| 16.5.1.2 | wWOCF + LOCF Imputation for the Pain Scores |
| 16.5.2 | Postoperative Consumption of Opioid Rescue Pain Medication |
| 16.5.3 | Overall Benefit of Analgesia Score Questionnaire |
| 16.5.4 | Subject Satisfaction with Postsurgical Pain Control |
| 16.5.5 | Sensitivity to Cold |
| | Predefined Treatment-Emergent Opioid-Related Adverse Events at |
| 16.5.6 | 72 Hours |
| 16.6.1 | Scheduled Bupivacaine Plasma Concentrations |
| 16.6.2 | Bupivacaine Plasma Pharmacokinetic Parameters |
| 16.6.3 | Unscheduled Bupivacaine Plasma Concentrations |
| 16.7.1.1 | Adverse Events (Part 1 of 2) |
| 16.7.1.2 | Adverse Events (Part 2 of 2) |
| 16.7.1.3 | Serious Adverse Events (Part 1 of 2) |
| 16.7.1.4 | Serious Adverse Events (Part 2 of 2) |
| 16.7.1.5 | Deaths |
| 16.8 | Height, Weight, and Vital Signs |
| 16.9 | Neurological Assessment |
| 16.10 | Physician's Satisfaction with Wound Healing |

Table 14.1.1.1 (Page x of Y) Subject Disposition (All Subjects)

| | LB | | All |
|---|---|---|---|
| | 266 mg | Placebo | Subjects |
| | (N=XX) | (N=XX) | (N=XX) |
| | <u>n (%)</u> | <u>n (%)</u> | <u>n (%)</u> |
| Safety Analysis Set [1] | 00(00.0) | 00(00.0) | 00(00.0) |
| Efficacy Analysis Set [2] | 00(00.0) | 00 (00.0) | 00 (00.0) |
| PK Analysis Set [3] | | NA | |
| Subjects Who Completed the Study | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Subjects Who Terminated Early | 00(00.0) | 00(00.0) | 00(00.0) |
| Reason for Early Termination | | | |
| Subject Death | 00(00.0) | 00(00.0) | 00(00.0) |
| Adverse Event | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Lack of Efficacy | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Lost to Follow-up | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Withdrawal by Subject | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Other Other | 00 (00.0) | 00 (00.0) | 00 (00.0) |

LB = liposome bupivacaine; PK = pharmacokinetic.

Reference: Listing 16.1.3.

<sup>[1]</sup> The safety analysis set includes all subjects who received study drug and is based on actual treatment received.

<sup>[2]</sup> The efficacy analysis set includes all subjects in the safety analysis set and is based on randomized treatment.

<sup>[3]</sup> The PK analysis set includes all subjects in the safety analysis set who received liposome bupivacaine and provided sufficient samples to allow for calculation of the PK parameters required for analysis.

Table 14.1.1.2 (Page x of Y)
Subject Disposition by Region and Site
(All Subjects)

| | | | LB | | All |
|---|---|---|---|---|---|
| | | | 266 mg | Placebo | Subjects |
| | | | (N=XX) | (N=XX) | (N=XX) |
| Region | Site | | <u>n (%)</u> | <u>n (%)</u> | <u>n (%)</u> |
| US | All Sites | Safety Analysis Set [1] | 00(00.0) | 00(00.0) | 00(00.0) |
| | | Efficacy Analysis Set [2] | 00(00.0) | 00(00.0) | 00(00.0) |
| | | PK Analysis Set [3] | | NA | |
| | | Subjects Who Completed the Study | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| | | Subjects Who Terminated Early | 00(00.0) | 00(00.0) | 00(00.0) |
| | | Reason for Early Termination | | | |
| | | Subject Death | 00(00.0) | 00(00.0) | 00(00.0) |
| | | Adverse Event | 00(00.0) | 00(00.0) | 00(00.0) |
| | | Lack of Efficacy | 00(00.0) | 00(00.0) | 00(00.0) |
| | | Lost to Follow-up | 00(00.0) | 00(00.0) | 00(00.0) |
| | | Withdrawal by Subject | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| | | Other | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| _ | <u>Etc</u> | | | | |

LB = liposome bupivacaine; PK = pharmacokinetic.

Reference: Listing 16.1.3.

<sup>[1]</sup> The safety analysis set includes all subjects who received study drug and is based on actual treatment received.

<sup>[2]</sup> The efficacy analysis set includes all subjects in the safety analysis set and is based on randomized treatment.

<sup>[3]</sup> The PK analysis set includes all subjects in the safety analysis set who received liposome bupivacaine and provided sufficient samples to allow for calculation of the PK parameters required for analysis.

Table 14.1.2 (Page x of Y)
Demographic and Baseline Characteristics
(Safety Analysis Set)

| | LB | | All |
|---|---|---|---|
| | 266 mg | Placebo | Subjects |
| | (N=XX) | (N=XX) | (N=XX) |
| | _ (1, 1111) | (11, 1111) | (11, 1111) |
| Age (years) | | | |
| N | 00 | 00 | 00 |
| Mean | 0.00 | 0.00 | 0.00 |
| SD | 00.00 | 00.00 | 00.00 |
| Median | 00 | 00 | 00 |
| Minimum, Maximum | 00, 00 | 00, 00 | 00,00 |
| , | , | , | , |
| Age Category | | | |
| <65 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| >=65 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Gender | | | |
| Male | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Female | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Ethnic Group | | | |
| Hispanic or Latino | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Not Hispanic or Latino | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Race [1] | | | |
| American Indian/Alaskan Native | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Asian | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Black or African American | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Native Hawaiian/Other Pacific Islander | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| White | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Other | , , | ` , | , |

LB = liposome bupivacaine.

Reference: Listing 16.2.

<sup>[1]</sup> Subjects may be counted in more than one category.

Table 14.1.2 (Page x of Y)
Demographic and Baseline Characteristics
(Safety Analysis Set)

| | LB | | All |
|------------------|-----------|-----------|-----------|
| | 266 mg | Placebo | Subjects |
| | _ (N=XX) | (N=XX) | (N=XX) |
| ASA Class | | | |
| 1 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| 2 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| 3 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Height (cm) | | | |
| n | 00 | 00 | 00 |
| Mean | 0.00 | 0.00 | 0.00 |
| SD | 00.00 | 00.00 | 00.00 |
| Median | 00 | 00 | 00 |
| Minimum, Maximum | 00,00 | 00,00 | 00,00 |
| Weight (kg) | | | |
| n | 00 | 00 | 00 |
| Mean | 0.00 | 0.00 | 0.00 |
| SD | 00.00 | 00.00 | 00.00 |
| Median | 00 | 00 | 00 |
| Minimum, Maximum | 00,00 | 00,00 | 00,00 |

ASA = American Society of Anesthesiologists; LB = liposome bupivacaine.

Reference: Listing 16.2.

<sup>[1]</sup> Subjects may be counted in more than one category.
Table 14.1.3.1 (Page x of Y)
Prior Medications
(Safety Analysis Set)

| ATC Class WHO-DD Preferred Term | LB<br>266 mg<br>(N=XX)<br><u>n (%)</u> | Placebo<br>(N=XX)<br><u>n (%)</u> | All Subjects (N=XX) n (%) |
|---|---|---|---|
| Any Prior Medication | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| ATC Class 1 Preferred Term 1 | 00 (00.0)<br>00 (00.0) | 00 (00.0)<br>00 (00.0) | 00 (00.0)<br>00 (00.0) |
| Preferred Term 2 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| ATC Class 2 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Preferred Term 3 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Preferred Term 4 Etc. | 00 (00.0) | 00 (00.0) | 00 (00.0) |

ATC = Anatomical Therapeutic Chemical classification system; LB = liposome bupivacaine; WHO-DD = World Health Organization Drug Dictionary

Note: Prior medications are defined as medication with a stop date/time prior to study drug administration. At each level of summation (overall, ATC class, and preferred term), subjects are only counted once.

Reference: Listing 16.3.4.

Table 14.1.3.2 (Page x of Y) Concomitant Medications (Safety Analysis Set)

| ATC Class WHO-DD Preferred Term | LB<br>266 mg<br>(N=XX)<br><u>n (%)</u> | Placebo<br>(N=XX)<br>n (%) | All Subjects (N=XX) n (%) |
|---|---|---|---|
| Any Prior Medication | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| ATC Class 1 Preferred Term 1 Preferred Term 2 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| ATC Class 2 Preferred Term 3 Preferred Term 4 Etc. | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| | 00 (00.0) | 00 (00.0) | 00 (00.0) |

ATC = Anatomical Therapeutic Chemical classification system; LB = liposome bupivacaine; WHO-DD = World Health Organization Drug Dictionary.

Note: Concomitant medications are defined as medications (other than rescue pain medication) taken on or after the start of study drug administration. This table does not include rescue pain medications.

At each level of summation (overall, ATC class, and preferred term), subjects are only counted once.

Reference: Listing 16.3.4.

Table 14.2.1.1 (Page x of Y) Study Drug Administration (Safety Analysis Set)

| | LB | |
|----------------------------------------|--------|---------|
| | 266 mg | Placebo |
| | (N=XX) | (N=XX) |
| Duration of Injection (min) | | |
| n | 00 | 00 |
| Mean | 0.00 | 0.00 |
| SD | 00.00 | 00.00 |
| Median | 00 | 00 |
| Minimum, Maximum | 00, 00 | 00,00 |
| Volume of Study Drug Administered (mL) | | |
| n | 00 | 00 |
| Mean | 0.00 | 0.00 |
| SD | 00.00 | 00.00 |
| Median | 00 | 00 |
| Minimum, Maximum | 00,00 | 00,00 |

LB = liposome bupivacaine.

Reference: Listing 16.4.1.

Table 14.2.1.2 (Page x of Y) Surgery (Efficacy Analysis Set)

| | LB | |
|---|---|---|
| | 266 mg | Placebo |
| | (N=XX) | (N=XX) |
| | <u> (11 222)</u> | <u>(11 /1/1)</u> |
| Duration of Surgery (min) | | |
| n | 00 | 00 |
| Mean | 0.00 | 0.00 |
| SD | 00.00 | 00.00 |
| Median | 00 | 00 |
| Minimum, Maximum | 00, 00 | 00,00 |
| Level of Index Nerve Injected | | |
| T3 | 00 (00.0) | 00 (00.0) |
| T4 | 00 (00.0) | 00 (00.0) |
| Etc. | ((())) | () |
| Location of Index Nerve Injected | | |
| Left | 00 (00.0) | 00 (00.0) |
| Right | 00 (00.0) | 00 (00.0) |
| At Least One Chest Tube Inserted | | |
| Yes | 00 (00.0) | 00 (00.0) |
| No | 00 (00.0) | 00 (00.0) |
| Time With Chest Tube(s) Inserted (min) [1] | | |
| n | 00 | 00 |
| Mean | 00.00 | 00.00 |
| SD | 00.000 | 00.000 |
| Median | 00.00 | 00.00 |
| Minimum, Maximum | 00.0, 00.0 | 00.0, 00.0 |
| | * | |

Time in ICU (hours)

| n | 00 | 00 |
|------------------|--------|-------|
| Mean | 0.00 | 0.00 |
| SD | 00.00 | 00.00 |
| Median | 00 | 00 |
| Minimum, Maximum | 00, 00 | 00,00 |

ICU = Intensive Care Unit; LB = liposome bupivacaine.

Reference: Listing 16.4.2 and 16.4.3.

<sup>[1]</sup> Since end of surgery. Only includes subjects who had at least one chest tube inserted.

## Table 14.2.2.1.1 (Page x of Y) AUC of NRS-R Pain Intensity Scores Through 72 Hours wWOCF + LOCF Imputation for the Pain Scores (Efficacy Analysis Set)

| | LB | |
|-------------------------------------|--------------|--------------|
| | 266 mg | Placebo |
| _ <u>Statistics</u> | (N=XX) | (N=XX) |
| n | 00 | 00 |
| Mean | 000.0 | 000.0 |
| SD | 00.00 | 00.00 |
| Median | 0000 | 0000 |
| Minimum, Maximum | 000, 000 | 000, 000 |
| LSM (Standard Error) [1] | 00.0 (00.00) | 00.0 (00.00) |
| LSM Difference (Standard Error) [2] | 00.0 (00.00) | , , |
| 95% CI for Difference [2] | 00.0, 00.0 | |
| P-value [2] | 0.0000 | |

AUC = area under the curve calculated using the trapezoidal method; CI = confidence interval; LB = liposome bupivacaine; LSM = least squares mean; NRS-R = numeric rating scale at rest.

Scores are based on a numeric rating scale where 0 = no pain and 10 = worst possible pain.

wWOCF + LOCF = imputation using the worst observation carried forward prior to the use of rescue medication within a medication window and last observation carried forward for missing values.

- [1] From an analysis of covariance with treatment and region (US and Europe) as main effects and the baseline NRS-R pain intensity score as a covariate.
- [2] Difference from placebo.

# Table 14.2.2.1.2 (Page x of Y) AUC of NRS-R Pain Intensity Scores Through 72 Hours by Region and Site wWOCF + LOCF Imputation for the Pain Scores (Efficacy Analysis Set)

| | | | LB<br>266 mg | Placebo |
|--------|-----------|------------------|--------------|----------|
| Region | Site | Statistics | (N=XX) | (N=XX) |
| US | All Sites | n | 00 | 00 |
| | | Mean | 0.000 | 0.000 |
| | | SD | 00.00 | 00.00 |
| | | Median | 0000 | 0000 |
| | | Minimum, Maximum | 000, 000 | 000, 000 |
| Etc. | Etc. | | | |

AUC = area under the curve calculated using the trapezoidal method; CI = confidence interval; LB = liposome bupivacaine; LSM = least squares mean; NRS-R = numeric rating scale at rest.

Scores are based on a numeric rating scale where 0 = no pain and 10 = worst possible pain.

wWOCF + LOCF = imputation using the worst observation carried forward prior to the use of rescue medication within a medication window and last observation carried forward for missing values.

Table 14.2.2.2 (Page x of Y)

Total Postoperative Consumption (mg) of Opioid Rescue Pain Medication Through 72 Hours

(Efficacy Analysis Set)

| Statistics | LB<br>266 mg<br>(N=XX) | Placebo<br>(N=XX) |
|-------------------------|------------------------|-------------------|
| n | 00 | 00 |
| Mean | 00.00 | 00.00 |
| Geometric Mean | 00.00 | 00.00 |
| SD | 00.000 | 00.000 |
| Median | 00.00 | 00.00 |
| Minimum, Maximum | 00.0, 00.0 | 00.0, 00.0 |
| Geometric LSM [1] | 00.00 | 00.00 |
| Geometric LSM Ratio [2] | 00.00 | |
| 95% CI for Ratio [2] | 00.00, 00.00 | |
| P-value [2] | 0.0000 | |

CI = confidence interval; LB = liposome bupivacaine; LSM = least squares mean.

If the total amount of opioid used was 0 mg, the value was set to the lesser of 1 mg or one half of the smallest total amount observed in the study prior to being transformed by the natural logarithm.

- [1] From an analysis of variance with treatment and region (US and Europe) as main effects on natural log transformed opioid amount. Results are presented in the original, non-transformed scale.
- [2] Geometric LSM Ratio is the anti-log LSM difference (LB/placebo).

Reference: Listing 16.5.2.

PCDOC #137836

26 February 2013

Pacira Pharmaceuticals, Inc. 402-C-322

Table 14.2.2.3 (Page x of Y) Time to First Opioid Rescue (Efficacy Analysis Set)

| | LB<br>266 mg<br>(N=XX) | Placebo<br>(N=XX) |
|---|---|---|
| Subjects Administered an Opioid Rescue [n (%)] | 00 (00.00) | 00 (00.00) |
| Censored Observations [n (%)] | 00 (00.00) | 00 (00.00) |
| Quartiles (hours) [1] | | |
| First Quartile (25% Administered an Opioid) | 000 | 000 |
| Median (50% Administered an Opioid) | 000 | 000 |
| Third Quartile (75% Administered an Opioid) | 000 | 000 |
| Minimum, Maximum | 00, 00* | 00, 00* |
| 95% CI of Median | (000, 000) | (000, 000) |
| P-value [2] | 0.0000 | |

<sup>\*</sup> indicates a censored observation.

Reference: Listing 16.5.2.

CI = confidence interval; LB = liposome bupivacaine.

<sup>[1]</sup> Kaplan-Meier estimates.

<sup>[2]</sup> Log-rank test with region (US and Europe) as a stratifying variable.

Table 14.2.2.4 (Page x of Y) NRS-R Pain Intensity Scores (Efficacy Analysis Set)

| | | LB | |
|---|---|---|---|
| | | 266 mg | Placebo |
| Time Point | Statistics | (N=XX) | (N=XX) |
| Baseline | n | 00 | 00 |
| | Mean | 0.000 | 0.000 |
| | SD | 00.00 | 00.00 |
| | Median | 0000 | 0000 |
| | Minimum, Maximum | 000, 000 | 000, 000 |
| First Request | n | 00 | 00 |
| 1 Hot Itoquest | Mean | 0.00 | 000.0 |
| | SD | 00.00 | 00.00 |
| | Median | 0000 | 0000 |
| | Minimum, Maximum | 000, 000 | 000, 000 |
| | LSM (Standard Error) [1] | 00.0 (00.00) | 00.0 (00.00) |
| | LSM Difference (Standard Error) [2] | 00.0 (00.00) | 00.0 (00.00) |
| | 95% CI for Difference [2] | 00.0, 00.0 | |
| | P-value [2] | 0.0000 | |
| 2 Hours | n | 00 | 00 |
| 2 Hours | Mean | 000.0 | 000.0 |
| | SD | 00.00 | 00.00 |
| | Median | 0000 | 0000 |
| | Minimum, Maximum | 000,000 | 000,000 |
| Etc. | IVIIIIIIIIIII, IVIAXIIIIIIII | 000, 000 | 000,000 |
| Lic. | | | |

CI = confidence interval; LB = liposome bupivacaine; LSM = least squares mean; NRS-R = numeric rating scale at rest. Scores are based on a numeric rating scale where <math>0 = no pain and 10 = worst possible pain.

Reference: Listing 16.5.1.1.

<sup>[1]</sup> From an analysis of covariance with treatment and region (US and Europe) as main effects and the baseline NRS-R pain intensity score as a covariate.

<sup>[2]</sup> Difference from placebo.

Table 14.2.2.5 (Page x of Y) NRS-A Pain Intensity Scores (Efficacy Analysis Set)

| | | LB | |
|---|---|---|---|
| | | 266 mg | Placebo |
| Time Point | Statistics | (N=XX) | (N=XX) |
| Baseline | n | 00 | 00 |
| | Mean | 0.000 | 0.000 |
| | SD | 00.00 | 00.00 |
| | Median | 0000 | 0000 |
| | Minimum, Maximum | 000, 000 | 000, 000 |
| First Request | n | 00 | 00 |
| 1 | Mean | 0.00 | 0.000 |
| | SD | 00.00 | 00.00 |
| | Median | 0000 | 0000 |
| | Minimum, Maximum | 000, 000 | 000, 000 |
| | LSM (Standard Error) [1] | 00.0 (00.00) | 00.0 (00.00) |
| | LSM Difference (Standard Error) [2] | 00.0 (00.00) | 00.0 (00.00) |
| | 95% CI for Difference [2] | 00.0, 00.0 | |
| | P-value [2] | 0.0000 | |
| 2 Hours | n | 00 | 00 |
| 2 110013 | Mean | 000.0 | 000.0 |
| | SD | 00.00 | 00.00 |
| | Median | 0000 | 0000 |
| | Minimum, Maximum | 000,000 | 000,000 |
| Etc. | ivininium, iviaximum | 000,000 | 000,000 |
| Lic. | | | |

CI = confidence interval; LB = liposome bupivacaine; LSM = least squares mean; NRS-A = numeric rating scale with activity. Scores are based on a numeric rating scale where <math>0 = no pain and 10 = worst possible pain.

Reference: Listing 16.5.1.1.

<sup>[1]</sup> From an analysis of covariance with treatment and region (US and Europe) as main effects and the baseline NRS-A pain intensity score as a covariate.

<sup>[2]</sup> Difference from placebo.

## Table 14.2.2.6 (Page x of Y) AUC of NRS-R Pain Intensity Scores Through 24, 36, 48, and 60 Hours wWOCF + LOCF Imputation for the Pain Scores (Efficacy Analysis Set)

| | LB | | |
|---|---|---|---|
| | | 266 mg | Placebo |
| Time Point | Statistics | (N=XX) | (N=XX) |
| 2411 | | 00 | 00 |
| 24 Hours | n | 00 | 00 |
| | Mean | 0.000 | 0.000 |
| | SD | 00.00 | 00.00 |
| | Median | 0000 | 0000 |
| | Minimum, Maximum | 000, 000 | 000, 000 |
| | LSM (Standard Error) [1] | 00.0 (00.00) | 00.0 (00.00) |
| | LSM Difference (Standard Error) [2] | 00.0 (00.00) | |
| | 95% CI for Difference [2] | 00.0, 00.0 | |
| | P-value [2] | 0.0000 | |
| 48 Hours | n | 00 | 00 |
| | Mean | 0.000 | 0.000 |
| | SD | 00.00 | 00.00 |
| | Median | 0000 | 0000 |
| | Minimum, Maximum | 000, 000 | 000, 000 |

Etc.

 $AUC = area \ under \ the \ curve \ calculated \ using \ the \ trapezoidal \ method; \ CI = confidence \ interval; \ LB = liposome \ bupivacaine;$ 

LSM = least squares mean; NRS-R = numeric rating scale at rest.

Scores are based on a numeric rating scale where 0 = no pain and 10 = worst possible pain.

wWOCF + LOCF = imputation using the worst observation carried forward prior to the use of rescue medication within a medication window and last observation carried forward for missing values.

- [1] From an analysis of covariance with treatment and region (US and Europe) as main effects and the baseline NRS-R pain intensity score as a covariate.
- [2] Difference from placebo.

## Table 14.2.2.7 (Page x of Y) AUC of NRS-R Pain Intensity Scores 24-48 and 48-72 Hours wWOCF + LOCF Imputation for the Pain Scores (Efficacy Analysis Set)

| | | LB | |
|---|---|---|---|
| | | 266 mg | Placebo |
| Time Point | Statistics | (N=XX) | (N=XX) |
| 24-48 Hours | n | 00 | 00 |
| | Mean | 0.000 | 0.000 |
| | SD | 00.00 | 00.00 |
| | Median | 0000 | 0000 |
| | Minimum, Maximum | 000, 000 | 000, 000 |
| | LSM (Standard Error) [1] | 00.0 (00.00) | 00.0 (00.00) |
| | LSM Difference (Standard Error) [2] | 00.0 (00.00) | , , |
| | 95% CI for Difference [2] | 00.0, 00.0 | |
| | P-value [2] | 0.0000 | |
| 48-72 Hours | n | 00 | 00 |
| | Mean | 0.000 | 0.000 |
| | SD | 00.00 | 00.00 |
| | Median | 0000 | 0000 |
| | Minimum, Maximum | 000,000 | 000, 000 |
| | LSM (Standard Error) [1] | 00.0 (00.00) | 00.0 (00.00) |
| | LSM Difference (Standard Error) [2] | 00.0 (00.00) | |
| | 95% CI for Difference [2] | 00.0, 00.0 | |
| | P-value [2] | 0.0000 | |

AUC = area under the curve calculated using the trapezoidal method; CI = confidence interval; LB = liposome bupivacaine; LSM = least squares mean; NRS-R = numeric rating scale at rest.

Scores are based on a numeric rating scale where 0 = no pain and 10 = worst possible pain.

wWOCF + LOCF = imputation using the worst observation carried forward prior to the use of rescue medication within a medication window and last observation carried forward for missing values.

- [1] From an analysis of covariance with treatment and region (US and Europe) as main effects and the baseline NRS-R pain intensity score as a covariate.
- [2] Difference from placebo.

Table 14.2.2.8 (Page x of Y)
Percentage of Subjects who are Pain Free at Each Time Point
(Efficacy Analysis Set)

| _ Time Point | LB<br>266 mg<br>(N=XX)<br><u>n/N (%)</u> | Placebo<br>(N=XX)<br>n/N (%) | <u>P-value [1]</u> |
|---|---|---|---|
| 1 Hour | 00/00 (00.0) | 00/00 (00.0) | 0.0000 |
| 2 Hours | 00/00 (00.0) | 00/00 (00.0) | 0.0000 |
| 4 Hours | 00/00 (00.0) | 00/00 (00.0) | 0.0000 |
| 8 Hours | 00/00 (00.0) | 00/00 (00.0) | 0.0000 |
| 12 Hours | 00/00 (00.0) | 00/00 (00.0) | 0.0000 |
| 24 Hours | 00/00 (00.0) | 00/00 (00.0) | 0.0000 |
| 36 Hours | 00/00 (00.0) | 00/00 (00.0) | 0.0000 |

Etc

Pain free is defined as a pain intensity score at rest of 0 or 1.

 $LB = liposome bupivacaine. \ n/N = Number of subjects with a pain score of 0 or 1/Number of subjects with a pain score at the time point.$ 

[1] P-value is from a chi-square test.

Reference: Listing 16.5.1.1.

Table 14.2.2.9 (Page x of Y)

Total Postoperative Consumption (mg) of Opioid Rescue Pain Medication Through 24, 36, 48, and 60 Hours (Efficacy Analysis Set)

| Time Point | Statistics | LB<br>266 mg<br>(N=XX) | Placebo<br>(N=XX) |
|---|---|---|---|
| 24 Hours | n | 00 | 00 |
| | Mean | 00.00 | 00.00 |
| | Geometric Mean | 00.00 | 00.00 |
| | SD | 00.000 | 00.000 |
| | Median | 00.00 | 00.00 |
| | Minimum, Maximum | 00.0, 00.0 | 00.0, 00.0 |
| | Geometric LSM [1] | 00.00 | 00.00 |
| | Geometric LSM Ratio [2] | 00.00 | |
| | 95% CI for Ratio [2] | 00.00, 00.00 | |
| | P-value [2] | 0.0000 | |
| E4- | = = | | |

Etc.

CI = confidence interval; LB = liposome bupivacaine; LSM = least squares mean.

If the total amount of opioid used was 0 mg, the value was set to the lesser of 1 mg or one half of the smallest total amount observed in the study prior to being transformed by the natural logarithm.

- [1] From an analysis of variance with treatment and region (US and Europe) as main effects on natural log transformed opioid amount. Results are presented in the original, non-transformed scale.
- [2] Geometric LSM ratio is the anti-log LSM difference (LB/placebo).

Reference: Listing 16.5.2.

Table 14.2.2.10 (Page x of Y)
Subjects Who Received Rescue Medication Through 72 Hours
(Efficacy Analysis Set)

| | LB<br>266 mg<br>(N=XX)<br>- n (%) | Placebo<br>(N=XX)<br>n (%) | <u>P-value [1]</u> |
|---|---|---|---|
| Received No Rescue Medication | 00 (00.0) | 00 (00.0) | 0.0000 |
| Received Only the First Rescue | 00 (00.0) | 00 (00.0) | 0.0000 |
| Received the First Rescue and a Second Opioid Rescue | 00 (00.0) | 00 (00.0) | 0.0000 |

LB = liposome bupivacaine.

[1] P-value is from a chi-square test

Reference: Listings 16.5.2.

Table 14.2.2.11 (Page x of Y)
Overall Benefit of Analgesia Score Questionnaire (Total Scores)
(Efficacy Analysis Set)

| | | LB | | |
|------------|------------------|----------|----------|-------------|
| | | 266 mg | Placebo | |
| Time Point | Statistics | (N=XX) | (N=XX) | P-value [1] |
| 24 Hours | _ | 00 | 00 | 0.0000 |
| 24 Hours | n<br>Mean | 000.0 | 000.0 | 0.0000 |
| | SD | 00.00 | 00.00 | |
| | Median | 0000 | 0000 | |
| | Minimum, Maximum | 000, 000 | 000, 000 | |
| 48 Hours | n | 00 | 00 | 0.0000 |
| | Mean | 000.0 | 0.000 | |
| | SD | 00.00 | 00.00 | |
| | Median | 0000 | 0000 | |
| | Minimum, Maximum | 000,000 | 000, 000 | |
| 72 Hours | n | 00 | 00 | 0.0000 |
| | Mean | 000.0 | 000.0 | |
| | SD | 00.00 | 00.00 | |
| | Median | 0000 | 0000 | |
| | Minimum, Maximum | 000, 000 | 000, 000 | |

LB = liposome bupivacaine.

Note: The lower the score, the greater the benefit of analgesia.

Reference: Listing 16.5.3.

<sup>[1]</sup> P-value is from a Wilcoxon Rank Sum test.

Table 14.2.2.12 (Page x of Y)
Subject Satisfaction with Postsurgical Pain Control
(Efficacy Analysis Set)

| | | LB | | |
|---|---|---|---|---|
| | | 266 mg | Placebo | |
| | | (N=XX) | (N=XX) | |
| Time Point | Assessment | n (%) | n (%) | P-value [1] |
| 72 Hours | Extremely Dissatisfied (1) | 00 (00.0) | 00(00.0) | 0.0000 |
| | Dissatisfied (2) | 00 (00.0) | 00(00.0) | |
| | Neither Satisfied nor Dissatisfied (3) | 00 (00.0) | 00(00.0) | |
| | Satisfied (4) | 00 (00.0) | 00 (00.0) | |
| | Extremely Satisfied (5) | 00 (00.0) | 00 (00.0) | |
| Day 12 | Extremely Dissatisfied (1) | 00 (00.0) | 00 (00.0) | 0.0000 |
| • | Dissatisfied (2) | 00 (00.0) | 00 (00.0) | |
| | Neither Satisfied nor Dissatisfied (3) | 00 (00.0) | 00 (00.0) | |
| | Satisfied (4) | 00 (00.0) | 00 (00.0) | |
| | Extremely Satisfied (5) | 00 (00.0) | 00 (00.0) | |
| Day 30 | Extremely Dissatisfied (1) | 00 (00.0) | 00 (00.0) | 0.0000 |
| • | Dissatisfied (2) | 00 (00.0) | 00 (00.0) | |
| | Neither Satisfied nor Dissatisfied (3) | 00 (00.0) | 00 (00.0) | |
| | Satisfied (4) | 00 (00.0) | 00 (00.0) | |
| | Extremely Satisfied (5) | 00 (00.0) | 00 (00.0) | |

LB = liposome bupivacaine.

Note: Percentages are based on number of subjects with a score at the time point.

Reference: Listing 16.5.4.

<sup>[1]</sup> P-value is from a Wilcoxon Rank Sum test.

Table 14.2.2.13 (Page x of Y)
Time to Sensitivity to Cold
(Safety Analysis Set)

| | LB | |
|-----------------------------------------------|------------|------------|
| | 266 mg | Placebo |
| | (N=XX) | (N=XX) |
| Subjects with Sensitivity to Cold [n (%)] | 00 (00.00) | 00 (00.00) |
| Censored Observations [n (%)] | 00 (00.00) | 00 (00.00) |
| Quartiles (hours) [1] | | |
| First Quartile (25% with Sensitivity to Cold) | 000 | 000 |
| Median (50% with Sensitivity to Cold) | 000 | 000 |
| Third Quartile (75% with Sensitivity to Cold) | 000 | 000 |
| Minimum, Maximum | 00, 00* | 00, 00* |
| 95% CI of Median | (000, 000) | (000, 000) |
| P-value [2] | 0.0000 | 0.0000 |

<sup>\*</sup> indicates a censored observation.

Reference: Listing 16.5.5.

CI = confidence interval; LB = liposome bupivacaine,

<sup>[1]</sup> Kaplan-Meier Estimates.

<sup>[2]</sup> Log-rank test with region (US and Europe) as a stratifying variable.

Table 14.2.2.14 (Page x of Y)
Incidence of Predefined Treatment-Emergent Opioid-Related Adverse Events
(Efficacy Analysis Set)

| <del>-</del> | LB<br>266 mg<br>(N=XX)<br><u>n (%)</u> | Placebo<br>(N=XX)<br>n (%) | <u>P-value [2]</u> |
|---|---|---|---|
| Subjects with at Least One Event | 00 (00.0) | 00 (00.0) | 0.0000 |
| Diffuse Pruritus | 00 (00.0) | 00 (00.0) | |
| Overt Respiratory Depression | 00 (00.0) | 00 (00.0) | |
| Urinary Retention [1] | 00 (00.0) | 00 (00.0) | |
| Constipation | 00 (00.0) | 00 (00.0) | |
| Sedation | 00 (00.0) | 00 (00.0) | |
| Confusion | 00 (00.0) | 00 (00.0) | |
| Delirium | 00 (00.0) | 00 (00.0) | |
| Vomiting | 00 (00.0) | 00 (00.0) | |
| Need for Antiemetic Medication | 00 (00.0) | 00 (00.0) | |

LB = liposome bupivacaine.

Reference: Listing 16.5.6.

<sup>[1]</sup> Urinary retention was measured by need for postsurgical bladder catheterization.

<sup>[2]</sup> P-value is from a chi-square test.

Table 14.2.3.1 (Page x of Y)
Bupivacaine Plasma Concentrations (ng/mL)
(PK Analysis Set)

| | | LB |
|---------------|-------------------|------------|
| | | 266 mg |
| _ Time Point | <u>Statistics</u> | (N=XX) |
| Baseline | n | 00 |
| | Mean | 000.00 |
| | SD | 0.000 |
| | %CV | 000.00 |
| | Median | 0.00 |
| | Minimum, Maximum | 00.0, 00.0 |
| 15 Minutes | n | 00 |
| | Mean | 000.00 |
| | SD | 0.000 |
| | %CV | 000.00 |
| | Median | 0.00 |
| | Minimum, Maximum | 00.0, 00.0 |
| 30 Minutes | n | 00 |
| | Mean | 000.00 |
| | SD | 0.000 |
| | %CV | 000.00 |
| | Median | 0.00 |
| | Minimum, Maximum | 00.0, 00.0 |
| _ <u>Etc.</u> | , | , |

LB = liposome bupivacaine.

Reference: Listing 16.6.1.

Table 14.2.3.2 (Page x of Y)
Bupivacaine Plasma Pharmacokinetic Parameters
(PK Analysis Set)

| | • | LB |
|---------------------|-------------------|--------------|
| | | 266 mg |
| <u>Parameter</u> | <u>Statistics</u> | (N=XX) |
| Cmax (ng/mL) | n | 00 |
| ommi (ng mz) | Mean | 000.00 0 |
| | SD | 0.0000 |
| | %CV | 000.00 |
| | Geometric Mean | 00.0 |
| | Median | 0.000 |
| | Minimum, Maximum | 00.00, 00.00 |
| Tmax (hours) | n | 00 |
| , | Mean | 000.00 0 |
| | SD | 0.0000 |
| | Median | 0.000 |
| | Minimum, Maximum | 00.00, 00.00 |
| AUC0-last (h*ng/mL) | n | 00 |
| ( 2 ) | Mean | 000.00 0 |
| | SD | 0.0000 |
| | %CV | 000.00 |
| | Geometric Mean | 0.00 |
| | Median | 0.000 |
| | Minimum, Maximum | 00.00, 00.00 |
| _ <u>Etc.</u> | | |

LB = liposome bupivacaine. Reference: Listing 16.6.2.

Programmer Note: The other parameters should be AUC0-inf (h\*ng/mL), and half-life (t1/2) (hours). %CV and geometric mean will not be shown for Tmax and half-life

Table 14.3.1.1 (Page x of Y)
Overview of Treatment-Emergent Adverse Events
(Safety Analysis Set)

| | LB<br>266 mg<br>(N=XX)<br>n (%) | Placebo<br>(N=XX)<br>n (%) | All Subjects (N=XX) n (%) |
|---|---|---|---|
| Subjects with at Least One TEAE | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Maximum Severity: Mild | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Maximum Severity: Moderate | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Maximum Severity: Severe | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| At Least One TEAE Related to Study Drug | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| At Least One Serious TEAE | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Subjects Discontinued Due to a TEAE | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Deaths on Study | 00 (00.0) | 00 (00.0) | 00 (00.0) |

LB = liposome bupivacaine; TEAE = treatment-emergent adverse event.

Table 14.3.1.2 (Page x of Y)
Incidence of Treatment-Emergent Adverse Events
(Safety Analysis Set)

| System Organ Class Preferred Term | LB<br>266 mg<br>(N=XX)<br><u>n (%)</u> | Placebo<br>(N=XX)<br>n (%) | All Subjects (N=XX) n (%) |
|---|---|---|---|
| Subjects with at Least One TEAE | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| System Organ Class 1 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Preferred Term 1 Preferred Term 2 | 00 (00.0)<br>00 (00.0) | 00 (00.0)<br>00 (00.0) | 00 (00.0)<br>00 (00.0) |
| System Organ Class 2 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Preferred Term 3 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Preferred Term 4 | 00 (00.0) | 00 (00.0) | 00 (00.0) |

Etc.

LB = liposome bupivacaine; TEAE = treatment-emergent adverse event.

At each level of summation (overall, system organ class, preferred term), subjects are only counted once.

Table 14.3.1.3 (Page x of Y)
Incidence of Study Drug Related Treatment-Emergent Adverse Events
(Safety Analysis Set)

| System Organ Class Preferred Term | LB<br>266 mg<br>(N=XX)<br><u>n (%)</u> | Placebo<br>(N=XX)<br>n (%) | All Subjects (N=XX) n (%) |
|---|---|---|---|
| Subjects with at Least One TEAE | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| System Organ Class 1 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Preferred Term 1 Preferred Term 2 | 00 (00.0)<br>00 (00.0) | 00 (00.0)<br>00 (00.0) | 00 (00.0)<br>00 (00.0) |
| System Organ Class 2 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Preferred Term 3 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Preferred Term 4 | 00 (00.0) | 00 (00.0) | 00 (00.0) |

Etc.

LB = liposome bupivacaine; TEAE = treatment-emergent adverse event.

At each level of summation (overall, system organ class, preferred term), subjects are only counted once.

Table 14.3.1.4 (Page x of Y)
Incidence of Treatment-Emergent Adverse Events by Severity
(Safety Analysis Set)

| | | LB | | | | | | All | |
|---|---|---|---|---|---|---|---|---|---|
| | | 266 mg | | | Placebo | | | Subjects | |
| | | (N = XX) | | | (N = XX) | | | (N = XX) | |
| System Organ Class | Mild | Moderate | Severe | Mild | Moderate | Severe | Mild | Moderate | Severe |
| Preferred Term | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subjects with at Least<br>One TEAE | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) |
| System Organ Class 1 | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) |
| Preferred Term 1 | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) |
| Preferred Term 2 | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) | 00 (00.00) |
| System Organ Class 2<br>Preferred Term 3<br>Preferred Term 4 | 00 (00.00)<br>00 (00.00)<br>00 (00.00) | 00 (00.00)<br>00 (00.00)<br>00 (00.00) | 00 (00.00)<br>00 (00.00)<br>00 (00.00) | 00 (00.00)<br>00 (00.00)<br>00 (00.00) | 00 (00.00)<br>00 (00.00)<br>00 (00.00) | 00 (00.00)<br>00 (00.00)<br>00 (00.00) | 00 (00.00)<br>00 (00.00)<br>00 (00.00) | 00 (00.00)<br>00 (00.00)<br>00 (00.00) | 00 (00.00)<br>00 (00.00)<br>00 (00.00) |

\_ ----

LB = liposome bupivacaine; TEAE = treatment-emergent adverse event.

At each level of summation (overall, system organ class, preferred term), subjects are only counted once using the highest severity.

Table 14.3.1.5 (Page x of Y)
Incidence of Serious Treatment-Emergent Adverse Events
(Safety Analysis Set)

| | LB | | All |
|---------------------------------|--------------|--------------|--------------|
| | 266 mg | Placebo | Subjects |
| System Organ Class | (N=XX) | (N=XX) | (N=XX) |
| Preferred Term | <u>n (%)</u> | <u>n (%)</u> | <u>n (%)</u> |
| Subjects with at Least One TEAE | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| System Organ Class 1 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Preferred Term 1 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Preferred Term 2 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| System Organ Class 2 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Preferred Term 3 | 00 (00.0) | 00 (00.0) | 00 (00.0) |
| Preferred Term 4 | 00 (00.0) | 00 (00.0) | 00 (00.0) |

Etc.

LB = liposome bupivacaine; TEAE = treatment-emergent adverse event.

At each level of summation (overall, system organ class, preferred term), subjects are only counted once.

Table 14.3.2.1 (Page x of Y) Vital Signs (Safety Analysis Set)

| | | | LB | |
|---|---|---|---|---|
| | | | 266 mg | Placebo |
| Parameter | Time Point | Statistics | (N=XX) | (N=XX) |
| | | | · | · |
| Heart Rate | Screening | n | 00 | 00 |
| | ū | Mean | 0.00 | 0.00 |
| | | SD | 00.00 | 00.00 |
| | | Median | 0.00 | 0.00 |
| | | Minimum, Maximum | 00, 00 | 00, 00 |
| | Baseline | n | 00 | 00 |
| | | Mean | 0.00 | 0.00 |
| | | SD | 00.00 | 00.00 |
| | | Median | 0.00 | 0.00 |
| | | Minimum, Maximum | 00, 00 | 00, 00 |
| | 1 Hour | n | 00 | 00 |
| | | Mean | 00.0 | 00.0 |
| | | SD | 00.00 | 00.00 |
| | | Median | 00.0 | 00.0 |
| | | Minimum, Maximum | 00, 00 | 00,00 |
| Etc. | Etc. | , | | |

LB = liposome bupivacaine.

Reference: Listing 16.8.

Table 14.3.2.2 (Page x of Y) Vital Signs Change from Baseline (Safety Analysis Set)

| | | | LB | |
|------------|------------|------------------|--------|---------|
| | | | 266 mg | Placebo |
| Parameter | Time Point | Statistics | (N=XX) | (N=XX) |
| Heart Rate | 1 Hour | n | 00 | 00 |
| | | Mean | 0.00 | 0.00 |
| | | SD | 00.00 | 00.00 |
| | | Median | 0.00 | 0.00 |
| | | Minimum, Maximum | 00, 00 | 00, 00 |
| | 12 Hours | n | 00 | 00 |
| | | Mean | 0.00 | 0.00 |
| | | SD | 00.00 | 00.00 |
| | | Median | 0.00 | 00.0 |
| | | Minimum, Maximum | 00, 00 | 00, 00 |
| | 24 Hours | n | 00 | 00 |
| | | Mean | 0.00 | 00.0 |
| | | SD | 00.00 | 00.00 |
| | | Median | 00.0 | 00.0 |
| | | Minimum, Maximum | 00, 00 | 00, 00 |
| Etc. | Etc. | | 23,00 | |

LB = liposome bupivacaine.

Reference: Listing 16.8.

Table 14.3.3 (Page x of Y) Neurological Assessment (Safety Analysis Set)

| _ Time Point | <u>Assessment</u> | LB<br>266 mg<br>(N=XX)<br><u>n/N (%)</u> | Placebo<br>(N=XX)<br>n/N (%) | All Subjects (N=XX) n/N (%) |
|---|---|---|---|---|
| Baseline | Oriented [1] At Least one of the Events Numbness [2] Metallic Taste in Mouth Problems with Hearing Problems with Vision Muscles Twitching | 00/00 (00.0)<br>00/00 (00.0) | 00/00 (00.0)<br>00/00 (00.0) | 00/00 (00.0)<br>00/00 (00.0) |
| 15 Minutes Etc. | Oriented [1] At Least one of the Events Numbness [2] Metallic Taste in Mouth Problems with Hearing Problems with Vision Muscles Twitching | 00/00 (00.0)<br>00/00 (00.0) | 00/00 (00.0)<br>00/00 (00.0) | 00/00 (00.0)<br>00/00 (00.0) |

LB = liposome bupivacaine. n/N = Number of subjects with a pain score of 0 or 1 / Number of subjects with a pain score at the time point.

Reference: Listing 16.9.

<sup>[1]</sup> The denominator does not include subjects who were not assessable at the time point.

<sup>[2]</sup> Numbness of the lips, the tongue, or around the mouth.

Table 14.3.4 (Page x of Y)
Physician's Satisfaction with Wound Healing
(Safety Analysis Set)

| Time Point | Assessment | LB<br>266 mg<br>(N=XX)<br>n (%) | Placebo<br>(N=XX)<br>n (%) | P-value [1] |
|---|---|---|---|---|
| 72 Hours | Extremely Dissatisfied (1) Dissatisfied (2) Neither Satisfied or Dissatisfied (3) Satisfied (4) Extremely Satisfied (5) | 00 (00.0)<br>00 (00.0)<br>00 (00.0)<br>00 (00.0)<br>00 (00.0) | 00 (00.0)<br>00 (00.0)<br>00 (00.0)<br>00 (00.0)<br>00 (00.0) | 0.0000 |
| Day 30 | Extremely Dissatisfied (1) Dissatisfied (2) Neither Satisfied or Dissatisfied (3) Satisfied (4) Extremely Satisfied (5) | 00 (00.0)<br>00 (00.0)<br>00 (00.0)<br>00 (00.0)<br>00 (00.0) | 00 (00.0)<br>00 (00.0)<br>00 (00.0)<br>00 (00.0)<br>00 (00.0) | 0.0000 |

LB = liposome bupivacaine.

Note: Percentages are based on number of subjects with a score at the time point.

Reference: Listing 16.10.

<sup>[1]</sup> P-value is from a Wilcoxon Rank Sum test.

#### LISTINGS

Listing 16.1.1 (Page x of Y) Eligibility

Treatment Group: YYY

| | | | | | | | Waiv | ver |
|---|---|---|---|---|---|---|---|---|
| | Date Informed | | | | | | | |
| | Consent Form | Randomization | Randomization | | Met Eligibility | Criteria Not | | |
| Subject ID | Signed | Date/Time | Number | Visit | Requirements? | Met | Granted? | Date |

Programmer note: Visit should be Registration, Screening, and Baseline. For Screening, the waiver questions should be blank.

#### Listing 16.1.2 (Page x of Y) Unblinding

| Treatment | Group: YYY | | | |
|---|---|---|---|---|
| Subject ID | Blind Broken? | Date of Unblinding | Reason | Person Who<br>Performed Unblinding |

Listing 16.1.3 (Page x of Y)
Subject Populations and Discontinuations

Treatment Group: YYY

| | | Subject Included In: | | | | | |
|---|---|---|---|---|---|---|---|
| | | | | | Date of Completion | | If Lost to |
| | Safety | Efficacy | PK | Complete the | or Early | Reason for Early | Follow-up, Date |
| Subject ID | Analysis Set [1] | Analysis Set [2] | Analysis Set [3] | Study? | Discontinuation | Discontinuation | of Last Contact |

PK = pharmacokinetic.

- [1] The safety analysis set includes all subjects who received study drug.
- [2] The efficacy analysis set includes all subjects in the safety analysis set.
- [3] The PK analysis set includes all subjects in the safety analysis set who received liposome bupivacaine and provided sufficient samples to allow for calculation of the PK parameters required for analysis.
### Listing 16.1.4 (Page x of Y) Hospital Discharge

| _ | Hospital Discharge | |
|------------|--------------------|------|
| Subject ID | Date | Time |

# Listing 16.2 (Page x of Y) Demographics and Baseline Characteristics

Treatment Group: YYY

| | | | | | | | ASA |
|---|---|---|---|---|---|---|---|
| Subject ID | Initials | Date of Birth | Age | Gender | Ethnicity | Race(s) | Class |

ASA = American Society of Anesthesiologists.

# Listing 16.3.1 (Page x of Y) Medical History Past Medical Findings or Surgical Procedures

Treatment Group: YYY

| Subject ID | Visit Date | Body System | Finding/<br>Procedure | Start Date | Currently Ongoing? |
|---|---|---|---|---|---|

Programmer note: Sort categories as on the CRFs, not alphabetically. If Other is checked for Body System then report as Other: specify.

Listing 16.3.2 (Page x of Y) Physical Examination

Treatment Group: YYY

Subject ID Performed? Date

# Listing 16.3.3 (Page x of Y) Electrocardiogram Recording (Holter Monitoring)

| Subject ID | Started? | Start Date | Start Time | Stop Date | Stop Time |
|------------|----------|------------|------------|-----------|-----------|

#### Listing 16.3.4

Prior and Concomitant Medications (Except for Protocol-Defined Rescue Pain Medications)

| Treatn | nent Group: YYY | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Anatomical Main Group/ | | | | | | | | _ |
| | Preferred Term / | Prior / | Reason for | AE Number | Start Date / | End Date / | | | |
| Subject ID | Verbatim Term | Concomitant | Use | or NA | Time | Time | Dose / Unit | Route | Frequency |

AE = adverse event; NA = Not applicable.

Prior medications are defined as medication with a stop date/time prior to study drug administration.

Concomitant medications are defined as medications (other than protocol-defined rescue pain medication) taken on or after the start of study drug administration.

Programmer note: If a subject has no medications, then put "NONE" in the 2nd column.

If the medication is Ongoing, then put "Ongoing" in the "End Date / Time" column.

Use formatted terms as much as possible. If you have to use codes, then add footnotes to explain the codes.

Listing 16.4.1 Study Drug Exposure

| | | | | Study | Drug Administration | |
|---|---|---|---|---|---|---|
| | Study Drug | Date | | | | Total |
| Subject ID | Administered? | Administered | Start Time | End Time | Duration (minutes) | Volume (mL) |

# Listing 16.4.2 Surgery

| | | Surgery | | Index Ner | | | |
|---|---|---|---|---|---|---|---|
| | | | | Duration | | | At Least One Chest |
| Subject ID | Date | Start Time | Stop Time | (minutes) | Level | Side | Tube Inserted? |

# Listing 16.4.3 Intensive Care Unit and Last Chest Tube Removal

Treatment Group: YYY

| | _ | ICU | | Last Chest Tube Removed | |
|---|---|---|---|---|---|
| Subject ID | Start Time | Time<br>Admitted | Time<br><u>Discharged</u> | <u>Date</u> | <u>Time</u> |

ICU = Intensive Care Unit.

# Listing 16.5.1.1 Pain Intensity Scores at Rest and with Activity

Treatment Group: YYY

<u>NRS-R</u> <u>NRS-A</u>

| | | Actual | Actual | | | | |
|---|---|---|---|---|---|---|---|
| Subject ID | Time Point | Date | Time | Actual Score | Imputed Score | Actual Score | Imputed Score |

NRS-R = numeric rating scale at rest; NRS-A = numeric rating scale with activity. Scores are based on a numeric rating scale where 0 = no pain and 10 = worst possible pain.

# Listing 16.5.1.2 AUC of NRS-R Pain Intensity Scores wWOCF + LOCF Imputation for the Pain Scores

Treatment Group: YYY

Time Interval
Subject ID (hours) AUC

AUC = area under the curve calculated using the trapezoidal method; NRS-R = numerical rating scale at rest.

Scores are based on a numeric rating scale where 0 = no pain and 10 = worst possible pain.

wWOCF + LOCF = imputation using the worst observation carried forward prior to the use of rescue medication within a medication window and last observation carried forward for missing values.

Programmer note: The Time Intervals should be 0-24, 0-36, 0-48, 0-72, 24-48, and 48-72.

# Listing 16.5.2 Postoperative Consumption of Opioid Rescue Pain Medication

Treatment Group: YYY

| | First or Second | | Date/Time | Hours from End | Amount Taken | | Converted | Cumulative |
|---|---|---|---|---|---|---|---|---|
| Subject ID | Rescue | Medication | Administered | of Surgery | (Units) | Route | Amount (mg) [1] | Amount (mg) |

[1] Opioids are converted to a morphine-equivalent amount.

Programmer note: If subject took no postoperative opioid pain medications, put 'NONE' in the 2nd column.

### Listing 16.5.3 Overall Benefit of Analgesia Score Questionnaire

| | | | Distress and Bother with [2]: | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | Satisfaction | |
| | | Date/Time of | Current Pain | | | | | | with Pain | |
| Subject ID | Time Point | Assessment | at Rest [1] | Vomiting | Itching | Sweating | Freezing | Dizziness | Treatment [2] | Total Score |

<sup>[1] 0 =</sup> Minimal Pain, 4 = Maximal imaginable pain.
[2] 0 = Not at all, 4 = Very much.

# Listing 16.5.4 Subject Satisfaction with Postsurgical Pain Control

| Subject ID Time Point | Date of Assessment | Time of<br>Assessment | Assessment |
|---|---|---|---|
|---|---|---|---|

### Listing 16.5.5 Sensitivity to Cold

| Treatment Group: YYY | | | | |
|---|---|---|---|---|
| Subject ID | Time Point | Date/Time of<br>Assessment | Sensitivity to Cold | - |

Listing 16.5.6
Predefined Treatment-Emergent Opioid-Related Adverse Events at 72 Hours

| | | | Overt | Urinary | | | | | | Need for |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Date of | Diffuse | Respiratory | Retention | | | | | | Antiemetic |
| ID | Assessment | Pruritus | Depression | [1] | Constipation | Sedation | Confusion | Delirium | Vomiting | Medication |

<sup>[1]</sup> Urinary retention was measured by need for postsurgical bladder catheterization.

# Listing 16.6.1 Scheduled Bupivacaine Plasma Concentrations

| | Dose Time | Date of | Time of | | Elapsed Time | Bupivacaine Plasma |
|---|---|---|---|---|---|---|
| Subject ID | [1] | Sample | Sample | Time Point | (hours) [2] | Concentration (ng/mL) |

<sup>[1]</sup> Dose time is the start time of study drug administration.

<sup>[2]</sup> Elapsed time is the time the sample was collected relative to the time of dose.

# Listing 16.6.2 Bupivacaine Plasma Pharmacokinetic Parameters

Treatment Group: YYY

### Listing 16.6.3 Unscheduled Bupivacaine Plasma Concentrations

| | Dose Time | Date of | Time of | Reason for | Elapsed Time | Bupivacaine Plasma |
|---|---|---|---|---|---|---|
| Subject ID | [1] | Sample | Sample | Collection | (hours) [2] | Concentration (ng/mL) |

<sup>[1]</sup> Dose time is the start time of study drug administration.

<sup>[2]</sup> Elapsed time is the time the sample was collected relative to the time of dose.

Listing 16.7.1.1 Adverse Events (Part 1 of 2)

Treatment Group: YYY

| | | | | Solicite | d From: | _ | | | |
|---|---|---|---|---|---|---|---|---|---|
| | SOC / | | | | | | | | |
| | Preferred Term / | Start Date / | End Date / | | | | | Relationship | |
| Subject ID | Verbatim Term | Time | Time | Neuro. [1] | ORAE[2] | Serious | Severity | to Study Drug | Outcome |

SOC = system organ class

<sup>\*</sup> Indicates that the event is not treatment-emergent.

<sup>[1]</sup> Neurological assessment.

<sup>[2]</sup> Predefined treatment-emergent opioid-related adverse events questionnaire.

Listing 16.7.1.2 Adverse Events (Part 2 of 2)

Treatment Group: YYY

| | | | | Action Taken with Subject | | | | |
|---|---|---|---|---|---|---|---|---|
| | SOC/ | | · | | | Non- | | |
| | Preferred Term / | Start Date / | End Date / | | | Pharmaceutical | Discontinued | |
| Subject ID | Verbatim Term | Time | Time | None | Medication | Therapy | from Study | Other |

SOC = system organ class.

<sup>\*</sup> Indicates that the event is not treatment-emergent.

Listing 16.7.1.3 Serious Adverse Events (Part 1 of 2)

Calinitad Ename.

Treatment Group: YYY

| | | | | Solicited | a From: | _ | | |
|---|---|---|---|---|---|---|---|---|
| | SOC / | | | | | | | |
| | Preferred Term / | Start Date / | End Date / | | | | Relationship | |
| Subject ID | Verbatim Term | Time | Time | Neuro. [1] | ORAE[2] | Severity | to Study Drug | Outcome |

SOC = system organ class.

<sup>\*</sup> Indicates that the event is not treatment-emergent.

<sup>[1]</sup> Neurological assessment.

<sup>[2]</sup> Predefined treatment-emergent opioid-related adverse events questionnaire.

### Listing 16.7.1.4 Serious Adverse Events (Part 2 of 2)

Treatment Group: YYY

| | | | | Action Taken with Subject | | | | |
|---|---|---|---|---|---|---|---|---|
| | SOC / | | | | | Non- | | |
| | Preferred Term / | Start Date / | End Date / | | | Pharmaceutical | Discontinued | |
| Subject ID | Verbatim Term | Time | Time | None | Medication | Therapy | from Study | Other |

SOC = system organ class.

<sup>\*</sup> Indicates that the event is not treatment-emergent.

Listing 16.7.1.5 Deaths

Treatment Group: YYY

Subject IDDatePrimary CauseAutopsyDate ofPart ofPrimary CausePerformed?Autopsy

Listing 16.8 Height, Weight, and Vital Signs

| | | | | | | | Blood Pressure (mmHg) | |
|---|---|---|---|---|---|---|---|---|
| | | | | | | Heart Rate | | |
| Subject ID | Time Point | Date | Time | Height (cm) | Weight (kg) | (bpm) | Systolic | Diastolic |

Listing 16.9 Neurological Assessment

| | | | | | | Metallic | Problems | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | Numbness | Taste in | with | Problems | Muscles |
| Subject ID | Time Point | Date | Time | Oriented | [1] | Mouth | Hearing | with Vision | Twitching |

<sup>[1]</sup> Numbness of the lips, the tongue, or around the mouth.

# Listing 16.10 Physician's Satisfaction with Wound Healing

Treatment Group: YYY

Date of Time of
Subject ID Time Point Assessment Assessment Assessment

### **Cardiac ECG Clinical Statistical Plan**

A Phase 3, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Assess the Efficacy and Safety of Intercostal Nerve Block with Liposome Bupivacaine in Subjects Undergoing Posterolateral Thoracotomy

Sponsor Reference: 402-C-322

#### **SPONSORED BY**

Pacira Pharmaceuticals, Inc. 10450 Science Center Drive San Diego, CA 92121 Tel: (858) 625-2424

This document is confidential.

**DATE**: 30Jul2013

V2

**By**: Joel Morganroth, M.D.

Chief Scientist, eResearchTechnology, Inc.

215 840 4961 (tel/cell)

610 527 0295 (fax)

JMorganroth@ert.com

Janyare

Signature:

## **TABLE OF CONTENTS**

| 1 | INTRODUCTION | 3 |
|-------|--------------------------------------------------|---|
| 1.1 | Objectives | 3 |
| 1.1.1 | Primary Objective | 3 |
| 1.1.2 | Secondary Objective | |
| 1.2 | Study Design | 4 |
| 1.3 | ECG Selection | 4 |
| 1.4 | Analysis of 12-Lead ECGs | 5 |
| 2 | ECG STATISTICAL PLAN | 6 |
| 2.1 | Subject Populations | 6 |
| 2.2 | Central Tendency Analysis | 6 |
| 2.3 | Outlier Analyses | 6 |
| 2.4 | Morphological Analysis | 7 |
| 3 | DEVIATIONS IN ANALYSIS FROM STATISTICAL PLAN AND | |
| | OTHER ISSUES | 8 |

#### 1 INTRODUCTION

Liposome bupivacaine was developed to extend pain relief with a single dose administration without the use of indwelling catheters and to decrease the requirement for supplemental opioid medications. It is indicated for use as an analgesic injected into the surgical site for postsurgical pain relief. This study explored the safety, efficacy, and pharmacokinetic (PK) profile of liposome bupivacaine when administered via a new route – intercostal nerve block.

Bupivacaine is one of the longer-acting local anesthetics, but even so it has a limited duration of action after local administration, usually reported as less than 8 hours. EXPAREL® (bupivacaine liposome injectable suspension; Pacira Pharmaceuticals, Inc., San Diego, California) consists of microscopic spherical, multivesicular liposomes (DepoFoam® drug delivery system), organized in a honeycomb-like structure comprising numerous non-concentric internal aqueous chambers containing a bupivacaine base at a concentration of 13.3 mg/mL. Each chamber is separated from adjacent chambers by lipid membranes. The lipids (phospholipids, cholesterol, and triglycerides) are naturally occurring or close analogs of endogenous lipids. Bupivacaine is slowly released from the DepoFoam particles by a complex mechanism involving reorganization of the barrier lipid membranes and subsequent diffusion of the drug over an extended period of time. A small amount of extra-liposomal bupivacaine (i.e., not bound within the DepoFoam particles) enables EXPAREL to have a similar onset of action to standard bupivacaine HCl.

EXPAREL was approved by the US FDA in 2011 for administration into the surgical site to produce postsurgical analysis. The active ingredient (bupivacaine) and inactive ingredient (DepoFoam) of EXPAREL are each contained, though separately, in FDA-approved products:

- Bupivacaine HCl solution, a well-characterized anesthetic/analgesic, with more than 35 years of use in the US.
- DepoFoam, a liposomal extended-release formulation contained in the marketed products DepoCyt(e)® (1999) and DepoDur® (2004). The form of DepoFoam used in each of the three products DepoCyt, DepoDur, and EXPAREL has a slightly different mixture of lipid components. However, unlike the other two products, EXPAREL employs a novel lipid excipient (dierucoylphosphatidylcholine [DEPC]) in its formulation.

#### 1.1 Objectives

#### 1.1.1 Primary Objective

The primary objective is to evaluate the efficacy of intercostal nerve block using liposome bupivacaine compared with placebo in subjects undergoing posterolateral thoracotomy.

### 1.1.2 Secondary Objectives

The secondary objectives are to evaluate additional efficacy parameters, assess the PK profile of liposome bupivacaine when administered as an intercostal nerve block, and further characterize the safety profile of liposome bupivacaine.

### 1.2 Study Design

This is a Phase 3, multicenter, randomized, double-blind, parallel-group, placebo-controlled study conducted to investigate the efficacy and safety of liposome bupivacaine (total of 266 mg in 20 mL) divided into three equal doses in three syringes of approximately 88 mg in 6.6 mL volume per nerve and administered to each of three nerve segments (index nerve, nerve above, and nerve below) compared with saline placebo nerve block. This study is to enroll 180 patients in up to 30 sites in the US and Europe.

After completing screening procedures, eligible subjects undergoing posterolateral thoracotomy will be randomized 1:1 to receive either liposome bupivacaine or placebo. Study drug will be administered after the posterolateral thoracotomy is completed (i.e., just prior to the surgical site closure).

This study will explore the safety and efficacy of liposome bupivacaine when administered via a new route – intercostal nerve block. Posterolateral thoracotomy model was selected as patients experience moderate to severe postsurgical pain that typically lasts for 2-3 days.

Exclusion criteria will include current or historical evidence of any clinically significant disease or condition, especially cardiovascular or neurological conditions that, in the opinion of the Investigator, may increase the risk of surgery or complicate the subject's postsurgical course or interfere with the determination of pain intensity related solely to the surgery.

### 1.3 ECG Selection

ECGs will be obtained by recording digital 12 lead ECGs on a Holter recorder (MORTARA H12+) started at baseline (approximately 1 hour prior to surgery) and will continue for a total of 72 hours. All subjects will have an ECG extracted at baseline and then post-treatment ECG(s) will be extracted at the determination of the  $T_{max}$  of bupivacaine for each study participant. Subjects who are treated with EXPAREL and have PK blood draws will have a single post-treatment ECG collected at actual  $T_{max}$ . Subjects who are treated with placebo or who do not have PK blood draws will have post-treatment ECGs extracted at both the mean and median  $T_{max}$ . The unblinded statistician will supply the mean and median  $T_{max}$  time points for these subjects based on the mean and median  $T_{max}$  observed in the EXPAREL treated subjects who have PK blood draws.

### 1.4 Analysis of 12-Lead ECGs

Digital 12-lead holter ECGs will be recorded using the Mortara Instrument Digital H12+TM ECG continuous recorder (Mortara Instrument, Inc., Milwaukee, Wisconsin), which will continuously record all 12 leads simultaneously from baseline (approximately 1 hour prior to surgery) and continue for 72 hours. The ECG signal will be recorded on compact flash memory cards provided to the sites. The subject's unique identification number and demographic information will be recorded for each flash card. Without knowledge of subject treatment assignment, the central laboratory, eResearchTechnology, Inc. (ERT; Philadelphia, PA, USA), will generate a 10-second, 12-lead digital ECG at baseline and at Tmax (see Section 1.3). If targeted ECG time points are artifactual and of poor quality, the central laboratory will capture analyzable 10-second ECGs as close as possible to the targeted time points.

Digital ECGs will be captured by the central laboratory and processed via its validated data management system, EXPERT. Interval duration measurements (IDMs) will first be obtained by trained analysts using the proprietary validated electronic caliper system applied on a computer screen utilizing the method of Global Median Beat. The Global Median Beat will be created by an algorithm, where one representative beat for each of the 12 leads is selected and superimposed, creating a single superimposed (Global Median) beat. Trained analysts will then review for correct interval duration measurement caliper placement and adjudicate the pre-placed algorithm calipers as necessary. A cardiologist will then verify the interval durations and perform the morphology analysis, noting any T-U wave complex that suggest an abnormal form compatible with an effect on cardiac repolarization.

On-screen measurements of heart rate (HR), PR, QRS, and QT interval durations will be performed and derived variables RR, QTcF, and QTcB will be calculated using the following formulae:

$$QTcB = QT/\sqrt{RR}$$

$$QTcF = QT/\sqrt{3}\sqrt{RR}$$

$$RR = 60/HR$$

Each fiducial point (onset of P wave, onset of Q wave, offset of S wave, and offset of T wave) will be marked. The original ECG waveform and such annotations will be saved separately in XML format for independent review.

Electrocardiogram changes in HR, RR, PR, QRS, QT, QTcF, and QTcB will be examined at T<sub>max</sub>.

#### 2 ECG STATISTICAL PLAN

### 2.1 Subject Populations

The ECG analysis will be performed on all enrolled subjects with at least one available pre-dose Day 1 baseline ECG and one post-dose ECG.

All data collected will be presented in data listings. Unscheduled ECG data, if available, will not be included in formal ECG analysis tables, but will be included in subject data listings.

Data from subjects excluded from an analysis population will be presented in the data listings, but will not be included in the calculation of summary statistics.

## 2.2 Central Tendency Analysis

The **baseline** ECG interval value will be obtained from the ECG extracted prior to study drug administration.

Descriptive statistics (e.g., frequency, percent, mean, standard deviation (SD), median, maximum and minimum) will be used to summarize the ECG variables and the corresponding changes from the baseline to the ECG(s) obtained at actual  $T_{max}$  when it is obtained, and when not, both the median and mean Tmax values will be used in each subject (see Section 1.3). This will provide a time point analysis which is detailed in the tables separately for placebo and liposome bupivacaine.

### 2.3 Outlier Analyses

An outlier analysis will supplement the central tendency analysis by determining if there are subjects who had an exaggerated effect on any ECG interval that would not be revealed in a mean change from baseline central tendency analysis.

Therefore, the data will be presented as the frequency and percent of subjects with each type of outlier. The following criteria ("study endpoints") are defined for this analysis ("new" means not present at baseline and becomes present on a post-dose ECG time point):

- Heart rate: A value for a subject is considered to be an outlier if the heart rate measurement at the post-dose time point is <50 bpm and the measure is at least a 25% decrease from the subject's baseline heart rate (i.e., a bradycardic event) or if the heart rate measurement at the post-dose time point is >100 bpm and the measure is at least a 25% increase from the baseline heart rate (i.e., a tachycardic event).
- <u>PR interval</u>: A value for a subject is considered to be an outlier if the PR interval at the post-dose time point is >200 ms and it is at least a 25% increase from the subject's baseline PR interval.

- QRS interval: A value for a subject is considered to be an outlier if the QRS interval at the post-dose time point is >100 ms and it is at least a 25% increase from the subject's baseline QRS interval.
- QT interval: A value for a subject is considered to be an outlier if the QT interval at the post-dose time point is >500 ms and the subject's baseline QT interval is  $\le 500$  ms.
- QTcF: A value for a subject is considered to be an outlier if the QTcF interval at the post-dose time point is >500 ms and the subject's baseline QTcF interval is ≤500 ms. Outlier values will also be presented if the QTcF interval at the post-dose time point is >480 ms when the subject's baseline QTcF interval is ≤480 ms and when the post-dose time point is >450 ms when the subject's baseline QTcF interval is ≤450 ms. In addition, the proportion of subjects with changes from baseline of >30-60 ms and >60 ms will be presented.
- QTcB: A value for a subject is considered to be an outlier if the QTcB interval at the post-dose time point is >500 ms and the subject's baseline QTcB interval is ≤500 ms. Outlier values will also be presented if the QTcB interval at the post-dose time point is >480 ms when the subject's baseline QTcB interval is ≤480 ms and when the post-dose time point is >450 ms when the subject's baseline QTcB interval is ≤450 ms. In addition, the proportion of subjects with changes from baseline of >30-60 ms and >60 ms will be presented.

The data will be presented by time point (actual  $T_{max}$ , mean  $T_{max}$  and median  $T_{max}$ ) separately for liposome bupivacaine and placebo.

A categorical or outlier analysis will be considered exploratory since the study was not powered to pick up unusual individual responses to the potential effects of drugs. Outlier analyses will produce data as the percentage of subjects in each treatment group that meet the criteria as defined for this analysis. All outliers will be summarized by treatment group on the basis of incidence rates. The outlier summary tables will include counts of subjects.

#### 2.4 Morphological Analysis

Morphological analyses will be performed with regard to the ECG waveform interpretation as defined by the central ECG laboratory's cardiologist. Changes from baseline to the post-dose ECG(s) will be done.

All findings will be presented in the ECG listings. New onset (presented as percentage of subjects meeting the new criteria) for the following variables will be detailed in the tables:

- Atrial fibrillation or flutter
- Second degree heart block,

- Third degree heart block,
- Complete right bundle branch block,
- Complete left bundle branch block,
- ST segment depression,
- ST segment elevation,
- T wave abnormalities (negative T waves only),
- Myocardial infarction pattern, and
- Any new abnormal U waves.

The data will be presented in the tables by time point (actual  $T_{max}$ , mean  $T_{max}$  and median  $T_{max}$ ) separately for the liposome bupivacaine and placebo groups as detailed above for the central tendency analyses.

# 3 DEVIATIONS IN ANALYSIS FROM STATISTICAL PLAN AND OTHER ISSUES

Deviations of the actual final statistical analysis from the statistical plan will be described and justified in the final report.